Compound No.: GTx-024

# GTx-024 as a Treatment for Stress Urinary Incontinence in Women: A Proof of Concept Study

Protocol G201001 Version 1.0 Confidential

Principal Investigator: Kenneth M. Peters, M.D.
Professor and Chair of Urology
Oakland University William Beaumont School of Medicine
3535 West 13 Mile Road, Suite 438
Royal Oak, MI 48073-6769
(248) 551-0387

E-mail: kmpeters@beaumont.edu

GTx Program Official: Michael DeSordi, BS, MBA Senior Director, Clinical Operations GTx, Inc. 175 Toyota Plaza, 7<sup>th</sup> Floor Memphis, TN 38103 Tel: (901) 261-3795 Fax: (901) 271-8679

E-mail: mdesordi@gtxinc.com

Version Number: 1.0 07 August 2015

Protocol Amendment Number: N/A

This template is adapted from the ICH guidance document E6 (Good Clinical Practice), Section 6.

GTx, Inc. SUI Protocol; Version 1.0 07 August 2015 

Compound No.: GTx-024

#### **CONFIDENTIALITY STATEMENT**

All information contained within this document are the joint property of GTx, Inc. and Oakland University William Beaumont School of Medicine (collectively, the Parties), and are considered confidential. Acceptance of this document constitutes the agreement by the Parties that no information contained herein may be divulged or disclosed by either Party to third parties without prior written approval of the other Party, except to the extent necessary to obtain informed consent from subjects who participate in this study or in connection with the reporting of serious adverse events as set forth in Section 9.2. Acceptance of this document by any recipient other than the Parties constitutes the agreement by such recipient that no information contained herein may be divulged or disclosed to third parties without prior written approval of GTx and Oakland University William Beaumont School of Medicine. Do not copy this protocol without the express written permission of GTx, Inc. and Oakland University William Beaumont School of Medicine.


Compound No.: GTx-024

#### STATEMENT OF COMPLIANCE

The study will be carried out in accordance with Good Clinical Practice (GCP) as required by the following:

 United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, and 21 CFR Part 312) ICH E6; 62 Federal Register 25691 (May 9, 1997)


Compound No.: GTx-024

#### **PROTOCOL SIGNATURE PAGE**

| Protocol Number: | G201001 | |
|---|---|---|
| Protocol Date: | 07 August 2015 | |
| Protocol Title: | GTx-024 as a Treatment for Stress<br>A Proof of Concept Study | Urinary Incontinence in Women: |
| SIGNATURE: | is Shoton | 08/07/15 |
| Sponsor | | Date |
| Mayzie Johnston V<br>Operations | .P Medical Affairs and Clinical | |
| Name and Title of | Sponsor Representative | |
| Principal Investiga | ator: | Date |
| Name of Principal | Investigator (Please Print) | |

The signature of the Sponsor Representative constitutes approval of this protocol. The signature of the Principal Investigator constitutes approval of this protocol and an assurance that this study will be conducted according to all requirements of this protocol and according to Good Clinical Practices (GCP).

Compound No.: GTx-024

### **TABLE OF CONTENTS**

| PROTOCOL SIGNATURE PAGE | 4 |
|---|---|
| TABLE OF CONTENTS | 5 |
| 1 PROTOCOL SUMMARY | 13 |
| 1.1 NAMES, AFFILIATIONS, AND ROLES OF CONTRIBUTING INDIVIDUALS | 18 |
| 2. INTRODUCTION: BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE | 20 |
| 2.1 BACKGROUND/RATIONALE | 20 |
| 2.2 RISKS ANALYSIS AND RISK ASSESSMENT | 26 |
| 2.2.1 POTENTIAL ANTICIPATED ADVERSE EVENTS | 26 |
| 2.2.2 STUDY RISKS | 29 |
| 3. OBJECTIVES | 30 |
| 3.1 PRIMARY OBJECTIVE | 30 |
| 3.2 SECONDARY OBJECTIVES | 30 |
| 3.3 STUDY ENDPOINTS | 32 |
| 4. METHODOLOGY | 33 |
| 4.1 STUDY DESIGN | 33 |
| 4.2 MEDICAL MONITORING | 33 |
| 5. STUDY ENROLLMENT AND WITHDRAWAL | 33 |
| 5.1 SUBJECT INCLUSION CRITERIA | 34 |
| 5.2 SUBJECT EXCLUSION CRITERIA | 34 |
| 5.3 STRATEGIES FOR RECRUITMENT, RETENTION, AND TO IMPROVE ADHERENCE INTERVENTION PROTOCOLS | E TO<br>35 |


Compound No.: GTx-024

| 5.4 | TREATMENT ASSESSMENT PROCEDURES | 35 |
|---|---|---|
| 5.4.1 | REASONS FOR WITHDRAWAL | 35 |
| 5.4.2 | EARLY TERMINATION OR SUSPENSION OF THE STUDY | 35 |
| 6. 8 | STUDY INTERVENTION/INVESTIGATIONAL PRODUCT | 36 |
| 6.1 | STUDY PRODUCT DESCRIPTION | 36 |
| 6.2 | ACQUISITION | 36 |
| 6.3 | FORMULATION, PACKAGING, AND LABELLING | 36 |
| 6.4 | PRODUCT STORAGE AND STABILITY | 36 |
| 6.5<br>INTEF | DOSAGE, PREPARATION, AND ADMINISTRATION OF STUDY RNEVTION/INVESTIGATIONAL PRODUCT | 36 |
| 6.6 | ACCOUNTABILITY PROCEDURES FOR THE STUDY INVESTIGATIONAL PRODUCT(S) | 36 |
| 6.7<br>INTEF | ASSESSMENT OF SUBJECT COMPLIANCE WITH STUDY RVENTION/INVESTIGATIONAL PRODUCT | 37 |
| 6.8 | CONCOMITANT MEDICATIONS/TREATMENTS | 38 |
| 7. \$ | STUDY SCHEDULE | 38 |
| 7.1 | STUDY VISITS | 38 |
| 7.2 | EARLY TERMINATION | 40 |
| 8. \$ | STUDY PROCEDURES/EVALUATIONS | 40 |
| 9. <i>A</i> | ASSESSMENT OF SAFETY | 43 |
| 9.1<br>PARA | METHODS AND TIMING FOR ASSESSING, RECORDING, AND ANALYZING SAFETY METERS | 43 |
| 9.1.1 | ADVERSE EVENTS | 43 |
| 9.1.2 | INTENSITY OF EVENT | 44 |
| 9.1.3 | DRUG – ADVERSE EVENT RELATIONSHIP | 44 |
| 9.1.4 | SERIOUS ADVERSE EVENTS | 45 |


Compound No.: GTx-024

| 9.2 | REPORTING PROCEDURES | 46 |
|---|---|---|
| 9.2.1 | SERIOUS ADVERSE EVENTS | 46 |
| 9.2.2 | REGULATORY REPORTING | 47 |
| 9.3 | TYPE AND DURATION OF FOLLOW-UP OF SUBJECTS AFTER ADVERSE EVENTS | 48 |
| 9.4 | HALTING RULES | 48 |
| 10. 5 | STATISTICAL CONSIDERATIONS | 49 |
| 10.1 | STATISTICAL METHODS | 49 |
| 11. C | QUALITY CONTROL AND QUALITY ASSURANCE | 51 |
| 12. E | THICS/PROTECTION OF HUMAN SUBJECTS | 52 |
| 12.1 | ETHICAL CONSIDERATIONS | 52 |
| 12.2 | INSTITUTIONAL REVIEW BOARD/ INDEPENDENT ETHICS COMMITTEE | 52 |
| 12.3 | PRE-STUDY DOCUMENTATION | 53 |
| 12.4 | INFORMED CONSENT PROCESS | 53 |
| 12.5 | SUBJECT CONFIDENTIALITY | 54 |
| 12.6 | PROTOCOL ADHERENCE | 54 |
| 12.7 | PERMISSION TO REVIEW SUBJECTS' SOURCE RECORDS | 54 |
| 12.8 | PROTOCOL AMENDMENTS | 54 |
| 12.9 | CHANGE IN INVESTIGATOR | 55 |
| 12.10 | STUDY DISCONTINUATION | 55 |
| 12.11 | INDEMNITY | 55 |
| 13. E | DATA HANDLING AND RECORD KEEPING | 55 |
| 13.1 | DATA CAPTURE METHODS | 56 |
| 13.1.1 | DATA COLLECTION | 56 |
| 13.2 | STUDY SITE RESPONSIBILITIES | 56 |


| | cocol: GTx-024 as a Treatment for Stress Urinary ontinence in Women: A Proof of Concept Study | Compound No.: GTx-024 | |
|---|---|---|---|
| 13.3 | CRF TIMING/REPORTS | | 56 |
| 13.4 | STUDY RECORDS RETENTION | | 56 |
| 13.5 | PROTOCOL DEVIATIONS | | 57 |
| 14. | PUBLICATION POLICY | | 58 |
| 15. | LITERATURE REFERENCES | | 59 |
| 1. | APPENDIX A: MESA URINARY QUESTIONI | NAIRE | 64 |
| (P | APPENDIX B: PATIENT GLOBAL IMPRESS<br>GI-S) SCALE AND PATIENT GLOBAL IMPRE<br>PROVEMENT (PGI-I) SCALE | | 67 |
| | APPENDIX C: URINARY DISTRESS INVENTONINENCE IMPACT QUESTIONNAIRE (III | • | 68 |
| 4. | APPENDIX D: FEMALE SEXUAL FUNCTION | N INDEX (FSFI) | 70 |
| 5. | APPENDIX E: VOIDING DIARY | | 76 |


Compound No.: GTx-024

#### LIST OF ABBREVIATIONS

AE Adverse Event

AMDC Adult Muscle Derived Cells

ALT Alanine Transaminase
AR Androgen Receptor

AR+/TNBC AR Positive, Triple Negative Breast Cancer

AST Aspartate Aminotransferase

BCRP Breast Cancer Resistance Protein

BMI Body Mass Index
°C Degrees Celsius
CB Clinical Benefit

CBC Complete Blood Count

CD-ROM Compact Disk Read Only Memory

CFR Code Of Federal Regulations

CR Complete Response

CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CTCAE Common Terminology Criteria For Adverse Events

DHEA Dehydroepiandrosterone

DHT Dihydrotestosterone

DSMB Data And Safety Monitoring Board

DXA Dual-Energy X-Ray Absorptiometry

EC Ethics Committee
ECG Electrocardiogram

ECOG Eastern Cooperative Oncology Group

EOS End of Study

CRF Case Report Form
EMG Electromyography
ER Estrogen Receptor


Compound No.: GTx-024

ER+BC Estrogen Receptor Positive Breast Cancer

°F Degrees Fahrenheit

FDA Food And Drug Administration
FSFI Female Sexual Function Index
FSH Follicle-stimulating hormone

GCP Good Clinical Practices

GGT Gamma-Glutamyl Transferase

GTx GTx, Inc.
GTx-024 Enobosarm

HBsAg Hepatitis B Surface Antigen
HDL High-Density Lipoprotein

HIV Human Immunodeficiency Virus
HRQOL Health Related Quality Of Life

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference On Harmonization

IEC Independent Ethics Committee

IIQ-7 Incontinence Impact Questionnaire
IMP Investigational Medicinal Product

IN Investigator Notification

IND Investigational New Drug Application

IRB Institutional Review Board

ISD Intrinsic Sphincter Deficiency

LBM Lean Body Mass

LDL Low-Density Lipoprotein

LUTS Lower Urinary Tract Symptoms

MESA Medical, Epidemiological And Social Aspects Of Aging

Mg Milligram

MMRM Mixed Model Repeat Measurement

MRI Magnetic Resonance Imaging

MUCP Maximum Urethral Closure Pressure


Compound No.: GTx-024

NA Not Applicable

NCI-CTCAE National Cancer Institute-Common Terminology Criteria For

Adverse Events

NOAEL No-Observable-Adverse-Effect-Levels

NSCLC Non-Small Cell Lung Cancer
PCOS Polycystic Ovarian Syndrome

Pgi-I Patient Global Impression Of Improvement Scale

Pgi-S Patient Global Impression Of Severity Scale

PFM Pelvic Floor Muscle

PFS Progression Free Survival

PI Principal Investigator

PO Per Os (Oral)

PrR Progesterone Receptor

PR Partial Response

PSA Prostate Specific Antigen

PT Physical Therapy
PVR Post Void Residual
QA Quality Assurance

QOL Quality of Life

RECIST Response Evaluation Criteria In Solid Tumors

SAE Serious Adverse Event SAP Statistical Analysis Plan

SARM Selective Androgen Receptor Modulator

SCP Stair Climb Power
SD Stable Disease

SHBG Sex Hormone Binding Globulin

SUI Stress Urinary Incontinence

SUSAR Suspected Unexpected Serious Adverse Reaction

TEAE Treatment Emergent Adverse Events

TNBC Triple Negative Breast Cancer

Compound No.: GTx-024

UA Urinalysis

UDI Urinary Distress Inventory

UI Urinary Incontinence

ULN Upper Limit of Normal

UNK Unknown

UPP Urethral Pressure Profile

US Ultrasound

UTI Urinary Tract Infection


Compound No.: GTx-024

### 1 PROTOCOL SUMMARY

| Title: | GTx-024 as a Treatment for Stress Urinary Incontinence in Women: A |
|---|---|
| | Proof of Concept Study |
| Sponsor: | GTx, Inc. |
| Indication: | Stress Urinary Incontinence (SUI) |
| Study Design: | This is a single site, single-arm, open-label proof of concept feasibility study. |
| Objectives: | Primary Objective Describe the effect of 12 weeks of treatment of GTx-024 on the number of stress incontinence episodes/day as assessed by the 3 day voiding diary. |
| | Secondary Objectives Describe the effect of 12 weeks of treatment of GTx-024 on the number of voids/day as assessed by the 3 day voiding diary. |
| | Describe the effect of 12 weeks of treatment of GTx-024 on urine volume per void as assessed by the 3 day voiding diary. |
| | Describe the effect of 12 weeks of treatment of GTx-024 on SUI as assessed by 24 hour pad weight test. |
| | Describe the effect of 12 weeks of treatment of GTx-024 on SUI as assessed by the Urethral Pressure Profile (UPP). |
| | Describe the effect of 12 weeks of treatment of GTx-024 on SUI as assessed by the Bladder Stress Test. |
| | Describe the effect of 12 weeks of treatment of GTx-024 on patient reported stress urinary incontinence symptoms as assessed by the MESA Urinary Questionnaire. |
| | Describe the effect of 12 weeks of treatment of GTx-024 on patient reported impression of stress urinary incontinence severity as assessed by the Patient Global Impression of Severity Scale (PGI-S) |
| | Describe the effect of 12 weeks of treatment of GTx-024 on patient reported impression of improvement as assessed by the Patient Global Impression of Improvement Scale (PGI-I). |
| | Describe the effect of 12 weeks of treatment of GTx-024 on patient reported urogenital distress as assessed by the Urinary Distress Inventory Questionnaire (UDI-6). |

Compound No.: GTx-024

Describe the effect of 12 weeks of treatment of GTx-024 on patient reported impact of urinary incontinence on daily life as assessed by the Incontinence Impact Questionnaire (IIQ-7).

Describe the effect of 12 weeks of treatment of GTx-024 on patient reported sexual function as indicated on the completion of the Female Sexual Function Index Questionnaire (FSFI).

Describe the effect of 12 weeks of treatment of GTx-024 on pelvic floor muscles as measured by MRI.

#### Safety objective:

To describe the safety profile of GTx-024 3 mg PO daily in subjects with SUI.

#### **Target Population:**

Adult postmenopausal women with SUI

**Subject Inclusion Criteria**: Subjects eligible for inclusion in this study must meet **all** of the following criteria:

- 1. Give voluntary, written and signed, informed consent
- 2. Female
- 3. Age 18 to 80 years old
- 4. Clinically confirmed as postmenopausal. Subjects must have undergone the onset of spontaneous, medically induced or surgical menopause prior to the start of this study. Postmenopausal is defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
- 5. SUI symptoms for at least 6 months duration
- 6. Predominant SUI (MESA questionnaire)
- 7. 24 hour pad weight >3 gms at baseline
- 8. At least 4, but no more than 15, SUI episodes on each day of the 3 day baseline voiding diary
- 9. Serum AST and ALT within normal limits
- 10. Total bilirubin within normal limits
- 11. Positive Bladder Stress Test
- 12.Subject agrees to not start any new treatment (medication or otherwise) that is known to affect lower urinary tract function throughout the treatment and follow up periods.
- 13. Subject agrees to maintain on a stable dose of any medication known to affect lower urinary tract function, including but not limited to anticholinergics, tricyclic antidepressants, or alpha-adrenergic blockers, throughout the treatment and follow-up period.

| Subject Exclusion Criteria: Subjects eligible for this study must not meet any of the following criteria: |
|---|
| <ol> <li>Pelvic floor physical therapy within the last 6 months</li> <li>History of pelvic radiation treatment</li> <li>History of urethral diverticula</li> <li>History of urethral sling, anterior prolapse repair, ureteral bulking agents and/or other SUI procedure or surgery</li> <li>Known vesicoureteral reflux, vaginal prolapse beyond the introitus, or other significant pelvic floor abnormalities</li> <li>Patient has urinary incontinence of neurogenic etiology</li> <li>Patient is morbidly obese (defined as 100 pounds over their ideal body weight, or body mass index 40 or greater)</li> <li>Chronic hepatitis</li> <li>Hepatic cirrhosis</li> <li>HIV and/or hepatitis A, B, or C</li> <li>Subjects taking systemic hormone products (excludes intravaginal application of estradiol topical/tablet agents and hormones delivered via vaginal rings)</li> <li>Subjects with a history of breast or endometrial cancer.</li> <li>Subjects with cerebrovascular disease, thromboembolic disorders, myocardial infarction, or angina.</li> <li>Subject with an entry measurement of &gt; 5 mm endometrial stripe thickness as measured by MRI.</li> </ol> |
| 15. Clinically confirmed urinary tract infection 16. Any other condition which per investigators' judgement may increase subject risk |
| 2 |
| 1 |
| 12 weeks |
| Up to 35 subjects. Each subject may complete up to 5 months of study |
| participation. |
| 6 months |
| GTx-024 has been tested as a treatment for muscle wasting associated |
| with cancer cachexia, but is not currently marketed. |
| Subjects will be instructed to take one 3 mg softgel capsule per day by |
| mouth, without regard to food intake. |

| Statistical | This is a proof of concept feasibility study, so no power calculation is |
|---|---|
| Considerations: | needed. Therefore, up to 35 subjects meeting inclusion/exclusion criteria will be recruited until 30 subjects have completed treatment. Descriptive statistics will be performed to explore changes in primary and secondary outcomes measures between baseline and end of treatment. The primary efficacy measure will be a reduction in the number of stress incontinence episodes/day. Secondary efficacy measures will include reduction in number of voids per day, volume of voids, 24 hour pad weight, responses to validated questionnaires, changes in UPP measures, changes in sexual function, and changes in pelvic floor muscles as measured by MRI. |
| | Safety will be determined by the number and type of adverse events reported during treatment. Various imputation methods may be explored. |
| Study | Participation in this study includes 5 in person study visits and two |
| Intervention/Treatment: | telephone and/or mailed questionnaire visits. Additional in person and/or |
| | telephone visits may be added as needed. |
| | Study subjects will receive 3 mg of GTx-024 orally daily. |

Compound No.: GTx-024

Table 1. Schedule of Measures.

| Table 1. 5 | Screening | Additional | Visit 1. | Visit 2. | Visit 3. | Visit 4. | Visit 5. | Visit 6. |
|---|---|---|---|---|---|---|---|---|
| | Visit<br>Days -21-0 | Screening<br>Days -21-0 | Baseline <sup>3</sup><br>Week 0 | Week 1± 3<br>days | Week 4 ± 3<br>days | Week 8 ± 3<br>days | Week 12 ± 3<br>days | Week 16 ±<br>7 days |
| | Clinic Visit | Clinic Visit | Clinic Visit | Phone Call | Clinic Visit | Clinic Visit | Clinic Visit | Phone Call<br>and Mail |
| Consent | х | | | | | | | |
| Inclusion/Exclusion | Х | | Х | | | | | |
| History | | | Х | | | | | |
| Interview/Vital<br>Signs | х | | Х | | Х | Х | х | |
| Height/Weight | х | | | | х | X | X | |
| 24 hour Pad Weight | Instruct | | х | | х | х | х | |
| 3 day Voiding Diary | Instruct | | X | | х | X | X | |
| Serum AST, ALT,<br>Total Bilirubin | х | | | | х | Х | х | |
| Serum FSH <sup>1</sup> , | Х | | | | | | | |
| CBC | | | Х | | | | Х | |
| UA Dipstick (with | Х | | Х | | | | Х | |
| culture as needed) | | | | | | | | |
| Lipid Panel | | | X | | | | Х | |
| Testosterone<br>Levels | | | Х | | | | X | |
| SHBG | | | Х | | | | Х | |
| UPP | | | Х | | | | х | |
| Pelvic MRI | | Х | | | | | Х | |
| Bladder Stress Test | х | | | | | | х | |
| Mammogram <sup>2</sup> | | х | | | | | | |
| Begin Daily⁴<br>Treatment | | | Х | | | | | |
| End Treatment | | | | | | | X | |
| Concomitant Meds | х | | X | X | X | X | X | X |
| Adverse Events | | | X | X | X | X | X | X |
| HIV, Hep A, B, C<br>Testing | х | | | | | | | |
| UDI-6; IIQ | | | X | | X | X | Х | Х |
| PGI-S | | | X | | X | X | X | X |
| MESA<br>Questionnaire | Х | | | | Х | Х | Х | Х |
| PGI-I | | | | | X | X | Х | Х |
| FSFI Questionnaire | | | x | | X | x | x | x |
| Bladder Scan PVR | | | X | | х | X | х | |
| Ciprofloxacin 500<br>mg po<br>(or equivalent) | | | Х | | | | Х | |
| Focused Physical<br>Exam | | | Х | | | | х | |

<sup>&</sup>lt;sup>1</sup> Age 18 to 80 years old is clinically confirmed as postmenopausal. Subjects must have undergone the onset of spontaneous, medically induced or surgical menopause prior to the start of this study. Postmenopausal is defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.

<sup>&</sup>lt;sup>2</sup> Mammogram within the last 6 months conducted outside the protocol may be utilized. Provided the data is available for assessment in this protocol, an additional mammogram will not be required.

<sup>&</sup>lt;sup>3</sup>Visit 1, Baseline, may not be completed until all results of screening tests have been evaluated.

<sup>&</sup>lt;sup>4</sup> After confirmation of meeting all eligibility criteria.

Compound No.: GTx-024

#### ROLES AND RESPONSIBILITIES

### 1.1 NAMES, AFFILIATIONS, AND ROLES OF CONTRIBUTING INDIVIDUALS

#### **Principal Investigator**

Kenneth M. Peters, M.D.
Professor and Chair of Urology
Oakland University William Beaumont School of Medicine
William Beaumont Hospital, Royal Oak
3535 W. 13 Mile Road Ste. 438
Royal Oak, MI 48073-6769
(248) 551-3637

E-mail: kmpeters@beaumont.edu

#### GTx, Inc.

Diane C. Young, M.D. Vice President, Chief Medical Officer GTx, Inc. 175 Toyota Plaza, 7<sup>th</sup> Floor Memphis, TN 38103 Tel: (901) 507-6948 Fax: (901) 271-8679

E-mail: dyoung@gtxinc.com

Michael DeSordi, BS, MBA Senior Director, Clinical Operations GTx, Inc. 175 Toyota Plaza, 7<sup>th</sup> Floor Memphis, TN 38103 Tel: (901) 261-3795

Fax: (901) 271-8679

E-mail: mdesordi@gtxinc.com

Mayzie Johnston, PharmD Vice President, Medical Affairs and Clinical Operations GTx, Inc. 175 Toyota Plaza, 7<sup>th</sup> Floor

Memphis, TN 38103 Tel: (901) 261-3858 Fax: (901) 271-8677

E-mail: mjohnston@gtxinc.com

Compound No.: GTx-024

Jeff Hesselberg, MBA Vice President, Regulatory Affairs, Corporate Quality & Drug Safety GTx, Inc. 175 Toyota Plaza, 7<sup>th</sup> Floor

Memphis TN 38103 Tel: (901) 523-9700 Fax: (901) 271-8707

E-mail: jhesselberg@gtxinc.com

Michael L. Hancock, MS Director, Biostatistics GTx, Inc. 175 Toyota Plaza, 7<sup>th</sup> Floor Memphis TN 38103 Tel: (901) 271-8700

Fax: (901) 271-8677

E-mail: mhancock@gtxinc.com

#### **Beaumont Hospital Clinical Research**

Larry T. Sirls, M.D., FACS
Professor of Urology
Oakland University William Beaumont School of Medicine
William Beaumont Hospital, Royal Oak
3535 W. 13 Mile Road Ste. 438
Royal Oak, MI 48073-6769
E-mail: lsirls@beaumont.edu

Kim Killinger, RN, MSN William Beaumont Hospital, Royal Oak 3535 W. 13 Mile Road Ste. 438 Royal Oak, MI 48073-6769 E-mail: KKillinger@beaumont.edu

Deborah Hasenau, RN, MS William Beaumont Hospital, Royal Oak 3535 W. 13 Mile Road Ste. 438 Royal Oak, MI 48073-6769

E-mail: Deborah.Hasenau@beaumont.edu

Compound No.: GTx-024

## 2. INTRODUCTION: BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE

#### 2.1 BACKGROUND/RATIONALE

Stress urinary incontinence (SUI), the involuntary leakage of urine during activities that increase abdominal pressure (e.g. coughing, sneezing, physical exercise), affects up to 35% of adult women (Luber, 2004). Urinary incontinence and pelvic floor disorders are major health problems for women especially as they age.

There are a variety of treatments that may be used to treat SUI in women (Rovner, 2004). Behavioral modification and pelvic floor physical therapy are common initial treatment approaches even though surgical procedures (e.g. sling; bladder neck suspension) are often ultimately the most effective. Biological and other materials for injection into the urethra have also been marketed for treating intrinsic sphincter deficiency (ISD), a cause of SUI symptoms. In a study of autologous fat injected into the urethral sphincter only 22% of patients improved compared to 21% after placebo injection (Lee, 2001). However, the injection of muscle derived stem cells (AMDC) is a promising new therapy for SUI currently being tested in clinical trials. In a dose escalation study of AMDC, injected into the urethral sphincter, all dose groups had significantly fewer diary stress leaks at 12 months, but only patients who received the highest dose of AMDC had statistically significant reduction in mean pad weight (Peters, 2014). Pharmacologic therapies for SUI also have been tested with varying results. In a study of duloxetine (a selective serotonin reuptake inhibitor), the median incontinence episode frequency decreased 41% in the placebo group compared to 54% receiving duloxetine 20 mg/day, 59% for duloxetine 40 mg/day, and 64% for duloxetine 80 mg/day (Norton, 2002). Dmochowski and colleagues also demonstrated a statistically significant reduction in incontinence episode frequency with duloxetine therapy compared with placebo (50% vs 27%, respectively) (Dmochowski, 2003).

Pelvic floor muscle relaxation has been found to correlate with lower urinary tract symptoms (LUTS). Muscles of the pelvic floor and lower urinary tract are crucial for supporting the pelvic organs and micturition, however damage to the muscles or lack of hormonal stimulation are thought to contribute to prolapse and urinary incontinence. As such, efforts have been made to improve pelvic floor muscle strength and function especially in post-reproductive and elderly women, to improve, if not cure, LUTS (specifically urinary incontinence, urinary frequency and nocturia). However, pelvic floor physical therapy (PT) is often less effective than more aggressive treatment such as surgery (Labrie, 2013). A prospective randomized trial of PT vs. surgery showed that 49% of women in the PT group crossed over to surgical treatment. Others have shown that after 3 to 15 years, 25 to 50% of women initially treated with physiotherapy have proceeded to surgery (Cammu, 2004; Lamers, 2007; B. K, Kvarstein, 2005). Yet, surgery is much more invasive and is associated with risk and complications (Brubaker

Compound No.: GTx-024

et al, 2011). Treatments with better outcomes than pelvic floor PT or those that augment the response to pelvic floor PT, are clearly needed. Androgen supplementation may be a novel treatment to augment pelvic floor muscle response and improve objective and subjective outcomes for SUI. Basic science literature indicates that smooth muscle cells in various female urogenital tissues have expressed androgen receptors (Berman, 2003) and that the levator ani and urethral sphincter, both containing large numbers of androgen receptors (Copas, 2001; Celayir, 2002), are sensitive to androgens (Nnodim, 1999; Nnodim, 2001).

In addition to the use of instruments to measure the efficacy of therapeutic approaches to SUI, MRI measurements of the pelvic floor have been utilized as tools to determine the impact on the supporting pelvic floor muscles (Tunn et al, 1999). Measurements of the levator hiatus, including the area, as well as, the anteroposterior and transverse diameters, have been demonstrated to be reproducibly measured and correlative with pelvic floor damage (Lammers et al., 2013). Similar measurements have been made to examine the recovery of levator ani muscle after vaginal delivery (Tunn et al, 1999). Therefore, MRI based measurements can provide for a non-invasive quantitative assessment of pelvic floor muscles and their potential response to therapeutic approaches with additional value to that provided by symptomatic assessments alone. MRI will also be used in this study to assess endometrial thickness at baseline. An endometrial stripe > 5 mm may exclude the subject from participating (Stanislavsky, Weerakkody, et al., 2015; Nakamura et al., 2014).

#### Androgen receptors in the pelvic floor/urethra

The para-urethral extracellular matrix is a target for sex steroid hormones, however the effects are not well known. Androgens stimulate collagen synthesis and inhibit degradation leading to increased collagen fibre compactness (Shin, 2005; Berger, 2005). Androgen receptors are densely expressed in both muscle and stromal cells of the levator ani muscle and fascia in women (Copas, 2001) and the levator ani muscle is considered to be one of the most androgen sensitive tissues in the body.

#### Impact of anabolic steroids

The effect of testoterone on urodynamic findings and histopathomorphology of the pelvic floor muscles has been studied in rat models of SUI. Testosterone was found to improve leak point pressures and significantly increase the size of myofibers in treated rats, suggesting that testosterone has both preventative and curative effects on rat models of SUI (Mammadov,2011). Since free testosterone levels were also higher in the treated group, there is potential for concerns regarding side effects of supplemental steroidal testosterone in women with SUI.

The anabolic effects of androgens in men have been widely studied, but less is known about the role and use of androgens in women. Prior studies have found that urinary levels of androgens were significantly higher in postmenopausal patients with SUI than in postmenopausal patients without incontinence (Jung, 2001). Furthermore, concentrations of androgen metabolites in urine of these patients were related positively

Compound No.: GTx-024

to the bladder neck descensus when measured by perineal ultrasound (a\_Bai, 2003). Aizawa K et al. and others have published data demonstrating that increases in muscle mass due to resistance training or exercise is due, at least in part, to increases in local androgen concentrations and expression of androgen-synthesizing enzymes (Aizawa K, 2011). These findings support the notion that pelvic floor muscle strengthening exercise improves SUI symptoms by increasing androgen levels locally. These and other studies suggest that androgens may play a substantial role in SUI and that androgen metabolites might be involved in the relaxation of bladder muscle (b\_Bai, 2003). This relaxation effect on the bladder may be related to the up regulation of nitric oxide synthase by androgens to produce more nitric oxide. The action of androgen on the lower urinary tract and pelvic floor is complex and may depend on anabolic effects, hormonal modulation, receptor expression, nitric oxide modulation, or combination of these factors (Ho MH, 2004).

Intriguing data come from studies conducted in women with polycystic ovarian syndrome (PCOS). PCOS is a hyper-androgenic disorder (>70 ng/dL compared to 15-50 ng/dL in normal pre-menopausal women) and clinical studies have demonstrated that PCOS can eliminate the increased risk for UI observed in obese women. Furthermore, obese women with PCOS have a similar prevalence of UI as those considered to have a normal body mass index (Montezuma T, 2011). In a separate study, none of the women with PCOS (18.6% with UI) suffered from UI compared to matched controls, even though pelvic floor muscle strength was not different (Antonio FI, 2013). These studies support the hypothesis that women with higher androgen levels, or potentially women treated with a selective androgen receptor modulator (SARM) will show improvements in UI symptoms.

#### Selective androgen receptor modulators

Although anabolic steroids may increase muscle mass and strength, lack of oral bioavailability and known potential risks have limited their use. Selective androgen receptor modulators (SARMS) have great potential to achieve similar benefits of anabolic steroid therapy (improved muscle mass, cholesterol/triglyceride levels, glucose metabolism, and bone density) with fewer adverse effects, such as hirsuitism and acne, in women.

SARMS may provide a new therapeutic option for pelvic floor and lower urinary tract disorders, as both testosterone and its more potent metabolite converted by 5-a reductase, dihydrotestosterone (DHT), have anabolic effects on muscle. The potential for SARMS as a treatment for SUI is strengthened by studies showing that urethral closure pressure is the factor most strongly associated with SUI (Delancey, 2007; Delancy, 2008). This finding is supported by both morphological and electromyographic (EMG) evidence. In imaging studies, the striated urethral sphincter has been found to be smaller in women with SUI compared to continent controls (Athanasiou, 1999; Morgan; 2009). In EMG studies, the striated urethral sphincters of women with SUI exhibit smaller EMG amplitudes and shorter motor-unit-potential durations, with more phases, than continent controls (Kenton, 2011; Takahashi, 2000), indicating primarily

Compound No.: GTx-024

myogenic changes. Furthermore, it is well accepted that pelvic floor muscle (PFM) rehabilitation is an effective treatment for SUI (Hay-Smith, 2009). PFM rehabilitation may be effective because it strengthens not only the pelvic floor but may also strengthen the striated urethral sphincter. This idea is supported by a recent publication that reported, based on ultrasound (US), a 12-week PFM exercise program produced a significant increase in the cross-sectional area of the urethra, at the level of the striated urethral sphincter, in middle-aged women (McLean, 2013). Because of limits in the resolution of US images, the authors were not able to determine which part of the urethra hypertrophied. The investigators suggested that PFM rehabilitation in older women with SUI could condition the striated urethral sphincter leading to measurable hypertrophy, observable on MRI.

In a later study, Madill extended the findings of the McLean group (Madill, 2014). Using MRI, they were able to differentiate between smooth and striated sphincter muscle layers and determined that changes occurred primarily in the striated urethral sphincter of older women. These findings suggest that not only does the striated urethral sphincter contract synergistically with PFMs during voluntary and automatic contractions [Nnodim, 1999; Nnodim, 2001; Celayir, 2002], but also that PFM rehabilitation stresses the striated urethral sphincter sufficiently to produce a muscular hypertrophy training effect (Madill, 2014).

Selective androgen receptor modulators (SARMS) are currently in development for patients with muscle wasting secondary to cancer diagnosis. This class of drugs has been shown to stimulate the growth of skeletal muscle, similar to traditional anabolic steroids, but without undesirable side effects. SARMS, such as GTx-024, are orally bioavailable and tissue-selective, whereas testosterone and other anabolic steroids also have limited oral bioavailability and are only available in transdermal and intramuscular formulations potentially leading to skin reactions and fluctuations in serum concentrations of testosterone. SARMS may exhibit the beneficial effects of anabolic agents without the known associated risks (Mohler, Bohl, 2009).

Recently utilizing an ovariectomized rat model to miminc SUI by disrupting urethral continence, investigators demonstrated that the use of a SARM (GSK2849466A) was able to increase urethral baseline pressure (UBP) and the amplitude of urethral responses during sneezing (AURS) by 64% and 74%, respectively, as compared with the vehicle control. Further, all of the rats (8/8) in the vehicle treated group experience fluid leakage during sneezing whereas only one of the rats (1/8) in the SARM treated group experience such leakage upon similar challenge. Histologically, the SARM treated animals had a reversal of the atrophy in urethral muscle observed in the control group. This preliminary in vivo study provides further support to the potential use of SARMs for the treatment of SUI. (Kadekawa et al, AUA Annual Meeting 2015, New Orleans, LA. PD27-11)

Compound No.: GTx-024

#### **Summary of GTx-024**

#### Preliminary studies related to stress urinary incontinence

Extensive clinical data related to the use of GTx-024 are described below; however. there are both pre-clinical and clinical data supporting the specific investigation of GTx-024 for the treatment of SUI. Among the preclinical findings are that GTx-024 has androgenic and anabolic activity in male and female rat models (Preclinical Reports n030105GTx024 and n112012.1). GTx-024 has consistently been observed to increase body weight, specifically muscle, in female rats. In a male rat model, with castrate levels of serum testosterone (similar to what might be expected in females), GTx-024 has the ability to induce hypertophy of the levator ani muscle to approximately 120% of an intact male. These studies together provide an approximation of the expected effect of GTx-024, since currently there are no data in female models regarding levator ani hypertrophy or stress urinary inconcentince (Preclinical Report n112012.1). In two phase 3 studies (G300504 and G300505), 3 mg daily GTx-024 results in a mild increase (approximately 1.7%) in lean body mass with no differential effect in males and females. Based upon these preclinical and clinical analyses, we anticipate significant growth/bulking of the levator ani in females with SUI, which may also result in improvements in associated symptoms, and are therefore the focus of the study outlined herein.

#### Ongoing and Completed Clinical Trials with GTx-024

The following Phase 1, 2, and 3 clinical trials have been completed or are ongoing with GTx-024.

- 1. Protocol G100401, a Phase 1 single ascending dose study in 96 healthy, young, male volunteers:
- 2. Protocol G100402, a Phase 1 multiple ascending dose study in 50 healthy, young, male volunteers, and 23 elderly male volunteers with truncal obesity;
- Protocol G100503, a Phase 1 single dose pharmacokinetic study to assess the
  effect of a dosage regimen that simulates a sustained release formulation to an
  immediate release formulation in 18 healthy, young male volunteers and 18
  postmenopausal women;
- 4. Protocol G100506, a Phase 1 single dose pharmacokinetic study to assess the relative bioavailability of a 3 mg hard shell capsule formulation to be used during continued clinical development and to assess the effect of food on the pharmacokinetics of the 3 mg softgel formulation in 27 healthy, young, male volunteers;
- 5. Protocol 006, a Phase 1 single dose and multiple dose pharmacokinetic study in 24 postmenopausal, Japanese women;
- 6. Protocol G200501, a Phase 2 study in 60 postmenopausal women and 60 elderly men to assess lean body mass and physical function;
- 7. Protocol 003, a Phase 1b study in 44 postmenopausal women;
- 8. Protocol G200502, a Phase 2b study in 159 men and postmenopausal women

Compound No.: GTx-024

- with cancer to assess lean body mass and physical function;
- 9. Protocol G100511, a Phase 1 study to assess the effect of severe renal impairment on the pharmacokinetics of GTx-024;
- 10. Protocol G100508, a Phase 1 study to assess the effect of mild and moderate hepatic impairment on the pharmacokinetics of GTx-024:
- 11. Protocol G100509, a Phase 1 mass balance study of GTx-024 in healthy volunteers;
- 12. Protocol G100507, a Phase 1 study to assess the pharmacokinetics and absolute oral bioavailability of GTx-024 in Caucasian and African American men and women;
- 13. Protocol G100510, a single-dose, randomized, double-blind, comparative, positive and placebo-controlled, four-period crossover Phase 1 study to define the electrocardiogram (ECG) effects of GTx-024, at therapeutic and supratherapeutic doses, in healthy male and female subjects: a thorough ECG trial;
- 14. Protocol G100512, a Phase 1 study to assess the effect of ketoconazole (Cytochrome P450, Family 3,Subfamily A [CYP3A4] inhibitor) on the pharmacokinetics of GTx-024;
- 15. Protocol G100513, a Phase 1 study to assess the effect of rifampin (CYP3A4 inducer) on the pharmacokinetics of GTx-024;
- 16. Protocol G100514, a Phase 1 study to assess the pharmacokinetic drug: drug interaction of GTx-024 and celecoxib (CYP2C9);
- 17. Protocol G100515, a Phase 1 study to assess the pharmacokinetic drug: drug interaction of GTx-024 and probenecid (UGT2B7);
- 18. Protocol G100516, a Phase 1 study to assess the pharmacokinetic drug: drug interaction of GTx-024 and rosuvastatin (breast cancer resistance protein [BCRP]):
- 19. Protocol G300504, a Phase 3 randomized, double-blind, placebo-controlled study of the effect of GTx-024 on muscle wasting in 321 subjects with non-small cell lung cancer receiving first line platinum plus a taxane chemotherapy;
- 20. Protocol G300505, a Phase 3 randomized, double-blind, placebo-controlled study of the effect of GTx-024 on muscle wasting in 320 subjects with non-small cell lung cancer receiving first line platinum plus a non-taxane chemotherapy;
- 21. Protocol G200801, an ongoing, Phase 2, open label study to examine AR status and the activity of GTx-024 hormonal therapy in 22 women with ER positive metastatic breast cancer who have previously responded to hormone therapy.
- 22. Protocol G200802, an ongoing, a Phase 2, open label, multi-center, multinational, randomized, parallel design study investigating the efficacy and safety of GTx-024 on metastatic or locally advanced ER+/AR+ Breast Cancer (BC) in Postmenopausal Women.
- 23. Protocol G200901, an ongoing, Phase 2, open label, multi-center, multinational study investigating the efficacy and safety of GTx-024 on advanced, Androgen Receptor-Positive Triple Negative Breast Cancer (AR+ TNBC)

Compound No.: GTx-024

#### 2.2 RISKS ANALYSIS AND RISK ASSESSMENT

#### 2.2.1 POTENTIAL ANTICIPATED ADVERSE EVENTS

An adverse event is any clinical event that impacts, or that has the potential to impact, the health or safety of a Clinical Study subject caused by or associated with the study device and/or testing. Assessment for potential adverse events will be ongoing throughout this trial.

The benefits of treatment may include improvement in the frequency, or severity of urine loss, and improvement in quality of life. Decreases in serum triglycerides, cholesterol, and body fat, and improvements in insulin resistance, lean body mass and physical endurance are also possible benefits.

Adverse event tables and serious adverse events discussed below and are presented separately by adverse events reported among healthy volunteers on a single trial of 86 days of GTx-024 3 mg versus placebo and those enrolled on cancer trials of at least 86 days exposure to GTx-024 3 mg or placebo.

# Adverse events reported among > 5% of GTx-024 3mg treated healthy subjects Percentage of subjects reporting a given adverse event at least once

| Primary System Organ Class | Preferred Term | GTx-024<br>N=24 | Placebo<br>N=24 |
|---|---|---|---|
| Gastrointestinal disorders | Diarrhea | 8.3 | 12.5 |
| | Dyspepsia | 8.3 | 8.3 |
| | Vomiting | 8.3 | 0.0 |
| General disorders and administration site conditions | Vessel puncture site bruise | 12.5 | 4.2 |
| | Fatigue | 8.3 | 8.3 |
| | Malaise | 8.3 | 0.0 |
| Infections and infestations | Herpes simplex | 8.3 | 0.0 |
| Injury, poisoning and procedural complications | Contusion | 8.3 | 4.2 |
| Investigations | Alanine aminotransferase increased | 20.8 | 0.0 |
| Musculoskeletal and connective tissue disorders | Back pain | 12.5 | 16.7 |

Compound No.: GTx-024

| Primary System Organ Class | Preferred Term | GTx-024<br>N=24 | |
|---|---|---|---|
| Nervous system disorders | Headache | 20.8 | 20.8 |
| | Dizziness | 12.5 | 4.2 |
| Respiratory, thoracic and mediastinal disorders | Pharyngolaryngeal pain | 12.5 | 12.5 |

No serious adverse events (SAEs) were reported on this trial.

These side effects are based on information obtained from a clinical study (G200501) administering GTx- 024 3 mg for 86 days in healthy subjects— elderly males and postmenopausal females. Studies suggest that side effects associated with the study drug resolve after GTx-024 is stopped.

#### Adverse events reported among > 5% of GTx-024 3 mg treated cancer subjects Percentage of subjects reporting a given adverse event at least once □

| Primary System Organ Class | Preferred Term | GTx-024<br>N=432 | Placebo<br>N=378 |
|---|---|---|---|
| Blood and lymphatic system disorders | Anemia | 34.7 | 34.7 |
| | Neutropenia | 18.3 | 23.3 |
| | Thrombocytopenia | 10.4 | 10.8 |
| | Leukopenia | 8.3 | 9.0 |
| Gastrointestinal disorders | Nausea | 34.7 | 34.9 |
| | Vomiting | 20.1 | 21.2 |
| | Constipation | 12.3 | 10.1 |
| | Diarrhea | 11.6 | 12.7 |
| | Abdominal pain | 5.1 | 3.7 |
| General disorders and administration site conditions | Fatigue | 15.7 | 16.7 |
| | Asthenia | 15.3 | 13.5 |
| | Disease progression | 11.8 | 16.7 |
| | Pyrexia | 10.2 | 9.8 |
| Infections and infestations | Pneumonia | 5.6 | 7.1 |
| Investigations | Blood creatinine increased | 8.1 | 5.0 |

Compound No.: GTx-024

| Primary System Organ Class | Preferred Term | GTx-024<br>N=432 | Placebo<br>N=378 |
|---|---|---|---|
| | Weight decreased | 6.0 | 4.8 |
| Metabolism and nutrition disorders | Decreased appetite | 10.6 | 14.8 |
| Musculoskeletal and connective tissue disorders | Arthralgia | 8.1 | 7.9 |
| | Pain in extremity | 5.6 | 4.2 |
| Nervous system disorders | Headache | 7.4 | 6.1 |
| | Peripheral sensory neuropathy | 5.8 | 3.4 |
| | Dizziness | 5.6 | 6.3 |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | 12.3 | 7.4 |
| | Cough | 9.5 | 9.3 |
| Skin and subcutaneous tissue disorders | Alopecia | 17.8 | 18.5 |

### Serious adverse events (SAEs) reported among > 2% of GTx-024 3 mg treated cancer subjects

Percentage of subjects reporting a given serious adverse event at least once

| Primary System Organ Class | Preferred Term | GTx-024<br>N=432 | Placebo<br>N=378 |
|---|---|---|---|
| Blood and lymphatic system disorders | Anemia | 4.2 | 3.7 |
| | Neutropenia | 3.2 | 3.7 |
| | Febrile neutropenia | 2.3 | 1.6 |
| Blood and lymphatic system disorders | Thrombocytopenia | 2.3 | 1.6 |
| General disorders and administration site conditions | Disease progression | 7.9 | 11.9 |
| Infections and infestations | Pneumonia | 3.5 | 3.2 |
| Neoplasms benign, malignant and unspecified (incl cysts and | Malignant neoplasm progression | 2.8 | 2.1 |

An AE that appears related to GTx-024 in clinical trials has been a dose-dependent, transient, asymptomatic increase in ALT. However, these increases were modest at doses up to 10 mg per day. Most of the subjects studied to date had ALT levels that

Compound No.: GTx-024

remained within normal limits. One subject was discontinued for an ALT > 3 times the ULN. The ALT levels returned to normal with continued exposure to GTx-024 in most cases and, further, in instances when dosing was not continued, levels returned to normal. No significant increases in total bilirubin, gamma glutamyl transferase, alkaline phosphatase, or lactate dehydrogenase have been observed in subjects with elevated ALT levels. Consistent with the effects of other orally administered anabolic agents, GTx-024 causes a dose dependent reduction in high-density lipoprotein (HDL), the clinical significance of which is unknown at this time. The proposed mechanism for reduction in HDL is due to stimulation of reverse cholesterol transport and increased HDL catabolism by hepatic lipase. Reductions in HDL are temporary and typically return to baseline 12 months after treatment initiation.

The effect of GTx-024 on a fetus has not been evaluated; therefore, the subjects in the current investigation will be post-menopausal.

#### 2.2.2 STUDY RISKS

#### **Study Procedures**

#### **Urethral catheterization**

Less Frequent (occurring more than 1%, but less than 10% of the time)

Discomfort

Mild cramping

Infection

Rare (occurring less than 1% of the time)

Bleeding

Urinary tract infection Inability to pass urine

Puncture of the bladder

Burning with urination

#### Antibiotic (a medicine to prevent infection)

Less Frequent (occurring more than 1% but less than 10% of the time)

Diarrhea

Nausea and vomiting

Cramping

Rare (occurring less than 1% of the time)

Headache

Itching

Rash

Allergic reaction

#### **Blood Drawing**

Most Frequent (occurring more than 10% of the time):

Pain

Bleeding

Compound No.: GTx-024

Bruising at the needle puncture site
Rare (occurring less than 1% of the time):
Blood clot
Infection
Feeling lightheaded
Fainting

#### Mammogram

Most Frequent (occurring more than 10% of the time):
Discomfort

#### **Gynecological Exam**

Rare (occurring less than 1% of the time):
Discomfort

#### Pelvic MRI

Rare (occurring less than 1% of the time):
Discomfort

#### 2.2.3 METHODS TO MINIMIZE RISK

Subjects will be monitored at each visit for changes since last visit and adverse effects of treatment. Since elevations in ALT are possible, serum liver function tests will be monitored during treatment. (Refer to Section 9.4 Halting Rules)

Subjects will receive a prophylactic antibiotic at visits where catheterization/UPP occur to decrease risk of urinary tract infection (UTI). Any infection will be appropriately treated.

#### 3. OBJECTIVES

#### 3.1 PRIMARY OBJECTIVE

1. Describe the effect of 12 weeks of treatment of GTx-024 on the number of stress incontinence episodes/day as assessed by the 3 day voiding diary.

#### 3.2 SECONDARY OBJECTIVES

- 1. Describe the effect of 12 weeks of treatment of GTx-024 on the frequency of voids/day as assessed by the 3 day voiding diary.
- 2. Describe the effect of 12 weeks of treatment of GTx-024 on urine volume per void as assessed by the 3 day voiding diary.


Compound No.: GTx-024

- 3. Describe the effect of 12 weeks of treatment of GTx-024 on SUI as assessed by 24 hour pad weight test.
- 4. Describe the effect of 12 weeks of treatment of GTx-024 on SUI as assessed by the Urethral Pressure Profile (UPP).
- 5. Describe the effect of 12 weeks of treatment of GTx-024 on SUI as assessed by the Bladder Stress Test.
- Describe the effect of 12 weeks of treatment of GTx-024 on patient reported stress urinary incontinence symptoms as assessed by the MESA Urinary Questionnaire.
- Describe the effect of 12 weeks of treatment of GTx-024 on patient reported impression of symptom severity as assessed by the Patient Global Impression of Severity Scale (PGI-S).
- 8. Describe the effect of 12 weeks of treatment of GTx-024 on patient reported impression of improvement as assessed by the Patient Global Impression of Improvement Scale (PGI-I).
- Describe the effect of 12 weeks of treatment of GTx-024 on patient reported urogenital distress as assessed by the Urinary Distress Inventory Questionnaire (UDI-6).
- 10. Describe the effect of 12 weeks of treatment of GTx-024 on patient reported impact of urinary incontinence on daily life as assessed by the Incontinence Impact Questionnaire (IIQ-7).
- 11. Describe the effect of 12 weeks of treatment of GTx-024 on patient reported sexual function as assessed by the Female Sexual Function Index Questionnaire (FSFI).
- 12. Describe the effect of 12 weeks of treatment of GTx-024 on pelvic floor muscles as measured by MRI.

Compound No.: GTx-024

#### 3.3 STUDY END POINTS

#### Primary end point

1. Change in frequency of daily stress urinary incontinence episodes from Baseline to Week 12.

#### Secondary end points

- 1. Change in frequency of daily voids from Baseline to Week 12.
- 2. Change in urine volume per void from Baseline to Week 12.
- 3. Change in 24 hour pad weight from Baseline to Week 12.
- 4. Change in maximum urethral closure pressure measurements from Baseline to Week 12.
- Change in urine leakage (yes/no) on the Bladder Stress Test from Baseline to Week 12 as assessed while (a) coughing, and/or (b) performing a Valsalva maneuver.
- 6. Change in total score on the stress incontinence section of the MESA Urinary Questionnaire from Baseline to Week 12.
- 7. Change in Patient Global Impression of Severity (PGI-S) Scale from Baseline to Week 12.
- 8. Patient Global Impression of Improvement (PGI-I) Scale at Week 12.
- Change in total score on the Urinary Distress Inventory (UDI-6) from Baseline to Week 12.
- 10. Change in total score on the Incontinence Impact Questionnaire (IIQ-7) from Baseline to Week 12.
- 11. Change in total score on the Female Sexual Function Index (FSFI) from Baseline to Week 12 as well as the change in subdomain scores: libido, arousal, lubrication, orgasm, satisfaction, and pain.
- 12. Change in pelvic floor muscles from Baseline to Week 12 as measured by MRI. Quantitative assessments may include the area of the levator hiatus, the anteroposterior and transverse diameters, and other relevant parameters.

Compound No.: GTx-024

#### 4. METHODOLOGY

#### 4.1 STUDY DESIGN

This is a single site, proof of concept feasibility study to describe the effect of GTx-024 3 mg in postmenopausal female subjects with SUI. Postmenopausal will be defined as clinically confirmed female subjects who have undergone the onset of spontaneous, medical or surgical menopause prior to the start of this study. Durability of treatment will also be explored by evaluating validated measures at 4 weeks after last dose. Up to 35 subjects will be enrolled in this study.

Institutional Review Board (IRB) approval from Beaumont's Human Investigations Committee will be obtained prior to beginning any study activity. Once IRB approval is obtained, potential participants will be identified from existing medical records, or physician or other referrals.

Potential subjects may be prescreened by telephone prior to the first in person study visit (initial screening visit). At the first in person study visit, subjects will be seen in the Urology Clinical Research space and informed consent will be obtained prior to any study activity. At Study Visit, 2, inclusion/exclusion criteria will be verified, study data will be collected, and consented participants may begin treatment.

Enrolled subjects will agree to maintain on a stable dose of any medication known to affect lower urinary tract function, including but not limited to anticholinergics, tricyclic antidepressants, or alpha-adrenergic blockers, throughout the treatment and follow-up period. Subjects enrolled in the study will agree to not start any new treatment (medication or otherwise) that is known to affect lower urinary tract function throughout the treatment and follow up periods. Subjects will also agree to refrain from performing any Kegal exercises and maintain current dietary habits throughout the treatment and follow up periods.

#### 4.2 MEDICAL MONITORING

A Medical Monitor will be responsible for monitoring the safety and data of this trial. The data that will be monitored include adverse events related to the study drug and procedures.

#### 5. STUDY ENROLLMENT AND WITHDRAWAL

#### 5.1 SUBJECT INCLUSION CRITERIA

**Subject Inclusion Criteria**: Subjects eligible for inclusion in this study must meet **all** of the following criteria:

- 1. Give voluntary, written and signed, informed consent
- 2. Female
- 3. Age 18 to 80 years old
- 4. Clinically confirmed as postmenopausal. Subjects must have undergone the onset of spontaneous, medically induced or surgical menopause prior to the start of this study. Postmenopausal is defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
- 5. SUI symptoms for at least 6 months duration
- 6. Predominant SUI (MESA questionnaire)
- 7. 24 hour pad weight >3 gms at baseline
- 8. At least 4, but no more than 15, SUI episodes on each day of the 3 day baseline voiding diary.
- 9. Serum AST and ALT within normal limits
- 10. Total bilirubin within normal limits
- 11. Positive Bladder Stress Test
- 12. Subject agrees to not start any new treatment (medication or otherwise) that is known to affect lower urinary tract function throughout the treatment and follow up periods.
- 13. Subject agrees to maintain on a stable dose of any medication known to affect lower urinary tract function, including but not limited to anticholinergics, tricyclic antidepressants, or alpha-adrenergic blockers, throughout the treatment and follow-up period.

#### 5.2 SUBJECT EXCLUSION CRITERIA

**Subject Exclusion Criteria**: Subjects eligible for this study must not meet any of the following criteria:

- 1. Pelvic floor physical therapy within the last 6 months
- 2. History of pelvic radiation treatment
- 3. History of urethral diverticula
- 4. History of urethral sling, anterior prolapse repair, ureteral bulking agents and/or other SUI procedure or surgery
- 5. Known vesicoureteral reflux, vaginal prolapse beyond the introitus, or other significant pelvic floor abnormalities
- 6. Patient has urinary incontinence of neurogenic etiology
- 7. Patient is morbidly obese (defined as 100 pounds over their ideal body weight, or body mass index 40 or greater)
- 8. Chronic hepatitis
- 9. Hepatic cirrhosis
- 10. HIV and/or hepatitis A, B, or C


Compound No.: GTx-024

- 11. Subjects taking systemic hormone products (excludes intravaginal application of estradiol topical/tablet agents and hormones delivered via vaginal rings)
- 12. Subjects with a history of breast or endometrial cancer.
- 13. Subjects with cerebrovascular disease, thromboembolic disorders, myocardial infarction, or angina.
- 14. Subject with an entry measurement of > 5 mm endometrial stripe thickness as measured by MRI.
- 15. Any other condition which per investigators' judgement may increase subject risk
- 16. Clinically confirmed urinary tract infection

## 5.3 STRATEGIES FOR RECRUITMENT, RETENTION, AND TO IMPROVE ADHERENCE TO INTERVENTION PROTOCOLS

Potential subjects will be identified from existing medical records, physician referrals, or recruited via advertisement or word of mouth. During initial telephone contact, patients' history will be reviewed for inclusion/exclusion criteria. Those subjects who initially qualify will be invited to an in person study visit (study visit 1).

#### 5.4 TREATMENT ASSIGNMENT PROCEDURES

All subjects enrolled in this study will receive a daily oral dose of GTx-024, 3 mg.

#### 5.4.1 REASONS FOR WITHDRAWAL

Subjects are free to withdraw from the study at any time for any reason.

In addition, subjects may be withdrawn from the study by the Principal Investigator (PI) in consultation with GTx, Inc. for reasons potentially including:

- Unable to tolerate study treatment (AE requiring permanent discontinuation of study treatment)
- AEs that require treatment with a prohibited medication or a procedure
- Development of any condition that may pose an additional risk to the subject or PI decision that this is in the best interest of the subject
- Study terminated by sponsor
- Subject unable to follow Investigators' instructions and comply with the study procedures
- Major protocol violation

The clinical study report will include reasons for all subject withdrawals from treatment and from the study as well as details relevant to violations of Study Prohibitions and Concomitant Therapy.

#### 5.4.2 EARLY TERMINATION OR SUSPENSION OF THE STUDY


Compound No.: GTx-024

Any decision to suspend enrollment or terminate the study will be made by the Sponsor, PI and, if appropriate, the local IRB. If a decision is made to terminate the study, subjects who have received treatment will be followed for up to 28 days.

#### 6. STUDY INTERVENTION/INVESTIGATIONAL PRODUCT

#### 6.1 STUDY PRODUCT DESCRIPTION

GTx-024 (enobosarm); United States Adopted Names Council official generic name) is an orally bioavailable nonsteroidal SARM with tissue-selective anabolic and androgenic pharmacologic activity (Dalton, 2011).

#### 6.2 ACQUISITION

GTx-024 3 mg Softgels (capsules) will be supplied by GTx, Inc.

#### 6.3 FORMULATION, PACKAGING, AND LABELLING

The drug product will be supplied as opaque, white to off-white, size 5, oval Softgel capsules containing 3 mg GTx-024. "GTx" will be imprinted in black ink on the outer shell of the capsule. The liquid Softgel fill is composed of GTx-024 dissolved in polyethylene glycol 400 (PEG400).

GTx-024 3 mg Softgels will be packaged in high density polyethylene (HDPE) bottles with induction seal and child-resistant closure. Each bottle will contain sufficient study drug for 35 days of dosing according to the study protocol. Each bottle of study drug will be labeled with dosing and storage instructions.

#### 6.4 PRODUCT STORAGE AND STABILITY

Recommended storage will be at controlled room temperature 15°C–25°C (59°F–77°F), with excursions permitted to 30°C (86°F), protected from moisture.

### 6.5 DOSAGE, PREPARATION, AND ADMINISTRATION OF STUDY INTERVENTION/INVESTIGATIONAL PRODUCT

One (1) GTx-024 3 mg Softgel capsule will be taken PO with water at approximately the same time each day, with or without food.

## 6.6 ACCOUNTABILITY PROCEDURES FOR THE STUDY INVESTIGATIONAL PRODUCT(S)

Compound No.: GTx-024

The Investigator is responsible for the correct storage of study medication according to GTx, Inc. recommendations. The study medication made available for this clinical trial must be used in accordance with the protocol and dispensed only under the supervision of the Investigator and documented sub-Investigators. The Investigator must maintain complete and accurate records, showing the receipt and disposition of all supplies of the study medication delivered by the GTx, Inc. authorized representative. These records must include a master record which lists the date of receipt of all study medication shipments, batch numbers, expiration date, and quantities received. In addition, a dispensing record which includes all quantities dispensed, identification of the subject to whom study medication was dispensed, the date of each dispensing, and the identification of the dispenser will also be maintained. The master dispensing records are separate from records kept for individual trial subjects.

It is the Investigator's responsibility to ensure that study medication used by trial subjects plus unused study medication equal the total amount received from the GTx, Inc. authorized representative. Damaged and/or contaminated packets must also be accounted for in the dispensing records. All discrepancies must be explained in writing. The study personnel responsible for study medication administration to the subject will record the date and time the initial treatment is given to the subject. In addition, the Drug Accountability case report form (CRF) will document any treatment interruptions or discontinuation.

## 6.7 ASSESSMENT OF SUBJECT COMPLIANCE WITH STUDY INTERVENTION/INVESTIGATIONAL PRODUCT

Subjects should be instructed to return all unused study medication and containers at each clinic visit during the clinical trial period so that drug accountability can be performed. The dispensing pharmacy is required to count all returned study capsules and record this on the proper CRF.

All study medication returned by subjects must be accounted for and verified by the study research nurse clinician and research pharmacist. After verification of all study medication, used packages and unused study medication will be returned to GTx, Inc., or authorized representative.

#### **Treatment Compliance**

Study subjects should be counseled on the need to meet 100% compliance with taking study drug. The investigator or designee should ensure that study subjects meet this goal throughout the study period. Compliance will be verified by the accounting of study drug at each in person visit after baseline. When study drug is administered at the research facility, it will be administered under the supervision of study personnel. Compliance with taking study drug will be monitored by the accounting of unused medication returned by the subject at visits. Compliance will be documented. If compliance is less than 80% or more than 120%, the Investigator or designee is to

Compound No.: GTx-024

counsel the subject and ensure steps are taken to improve compliance. Subjects who are less than 80% or more than 120% compliant with the dosage regimen for any two consecutive visit periods during the study may be withdrawn from the study.

#### 6.8 CONCOMITANT MEDICATIONS/TREATMENTS

Forbidden medications and treatments during the study duration include:

- Systemic hormonal products including but not limited to estrogens, progestins, testosterone, methyltestosterone, oxandrolone (Oxandrin®), oxymetholone, danazol, fluoxymesterone (Halotestin®), other androgenic compounds, including herbals. Intravaginal application of estradiol topical/tablet agents and hormones delivered via vaginal ring are allowed.
- Treatment with any investigational agent within 6 months before the first dose of study treatment;

Previous and Concomitant Medication (Drugs and Therapies)

The Investigator or designee must record the use of previous (all medication taken within 30 days prior to Screening (Visit 1) and current concomitant treatment, both drug and non-drug therapies, prescribed and over-the-counter and all alternative medicines, in the CRFs. This also includes drugs used on a chronic and as-needed basis. Subjects must be instructed not to start any new medication, both prescribed and over-the-counter, without consulting the Investigator, unless the new medication is required for emergency use. Subjects must be instructed to notify the Investigator immediately if medications were required for emergency use.

#### 7. STUDY SCHEDULE

#### 7.1 STUDY VISITS

Each subject may complete up to 5 months of study participation.

Screening Visit, Days -21-0

The study will be explained in detail and adequate time will be allowed for answering potential subjects questions prior to signing the IRB approved informed consent document. Informed consent will be obtained from those volunteers meeting initial inclusion/exclusion criteria and expressing willingness to participate prior to conducting any further study tests or measures.

Once informed consent is obtained, a detailed interview with vital signs will be conducted to further review for inclusion/exclusion criteria. A subject number will be assigned. Height and weight will be measured. Subjects will complete the MESA questionnaire to assess incontinence type (stress, urge, or mixed). If urinary incontinence type is stress predominant, then the subject will be instructed to complete a 24 hour pad weight and 3 day voiding diary prior to the next study visit. A bladder

Compound No.: GTx-024

stress test will be done to confirm SUI. Lab tests will also be drawn at this visit as outlined in Table I. A baseline urinalysis will be obtained. Concomitant medications will also be assessed and recorded.

#### Additional Screening, Days -21-0

If the subject has qualified for the study during the Screening visit, the following procedures will be performed between Screening Visit and Visit 1. Mammogram, if not done within the last 6 months, will be performed. Pelvic MRI will be performed

#### Study Visit 1: Week 0, Clinic Visit

Subjects still meeting inclusion/exclusion criteria after all Screening study measures have been completed and reviewed will return for Visit 1 where the 24 hour pad weight and 3 day voiding diary will be collected and reviewed. An interview with vital signs will be conducted. A detailed medical history will be taken, including past gynecological and obstetric history (gravida, para, prior abortions and deliveries) and a focused physical exam, including standard gynecological pelvic exam and skin assessment, will be done. Urine dipstick will be done and PVR will be measured. If subject still meets inclusion/exclusion criteria, UPP will be performed. A dose of Ciprofloxacin or equivalent will be given prophylactically to prevent bladder infection. Serum lab tests consisting of a CBC, lipid panel and testosterone level will be drawn.Questionnaires (UDI-6, IIQ, FSFI, and PGI-S) will also be completed at this visit. Concomitant medications and adverse events, will be assessed and recorded. A baseline MRI measurement will be scheduled and/or completed prior to receiving study drug.

Subjects who meet all the inclusion and none of the exclusion criteria will receive study drug. Study drug will be packaged in bottles. Each study drug bottle will be preprinted with a Medication ID number. The Medication ID number assigned to the subject will be noted in the case report form (CRF) for study drug.

The first dose of study drug will be taken during this visit if the subject meets all criteria for enrollment. A one month supply of study drug (35 count bottles) will be dispensed with administration instructions.

#### Study Visit 2: Week 1, Phone Call

Approximately 1 week after beginning treatment, subjects will be contacted by phone to assess for concomitant meds and adverse events. Subjects will also be instructed to complete a 24 hour pad weight and 3 day voiding diary within the week preceding their next study visit.

#### Study Visit 3: Week 4, Clinic Visit

Approximately 4 weeks after beginning treatment, subjects will return to the clinical research office for an in person visit. An interview with vital signs will be conducted. Height and weight and PVR will be measured. Pad weights will be measured, and the 3 day voiding diary will be collected and reviewed. Blood will also be drawn to measure serum AST, ALT, and total bilirubin. Questionnaires will also be completed, and

Compound No.: GTx-024

concomitant meds and adverse events, including any vaginal bleeding, discharge, infections and/or spotting, will be assessed and recorded. Subjects will also be instructed to complete a 24 hour pad weight and 3 day voiding diary in the week preceding their next study visit. A 30 day supply of study drug will be dispensed with administration instructions.

#### Study Visit 4: Week 8, Clinic Visit

Approximately 8 weeks after beginning treatment, subjects will return to the clinical research office for an in person visit. An interview and vital signs will be conducted. Height and weight and PVR will be measured. Pad weights will be measured, and the 3 day voiding diary will be collected and reviewed. Blood will also be drawn to measure serum AST, ALT, and total bilirubin. Questionnaires will also be completed and concomitant meds and adverse events including any vaginal bleeding, discharge, infections and/or spotting,will be assessed and recorded. Subjects will also be instructed to complete a 24 hour pad weight and 3 day voiding diary in the week preceding their next study visit. A 30 day supply of study drug will be dispensed with administration instructions.

#### Study Visit 5: Week 12, Clinic Visit

Approximately 12 weeks after beginning treatment, subjects will return to the clinical research office for an in person visit. An interview with vital signs will be conducted. A focused physical exam will be done. Gynecological pelvic exam will only be done at this visit if clinically indicated. Urine dipstick will be done and PVR will be measured Height and weight will be measured. 24 hour pad weights and 3 day voiding diaries will be collected/reviewed. Blood will also be drawn to measure laboratory values as outlined in Table 1. UPP,Bladder Stress Test, and MRI will be performed at end of treatment, questionnaires will be administered, and concomitant medications/adverse events will be assessed and recorded. All study medication will be collected and accounted for.

Study Visit 6: Week 16, Telephone/mailed questionnaire visit Approximately 4 weeks after study drug treatment has ended, subjects will be contacted by phone to assess for concomitant meds and adverse events. Subjects will also be instructed to complete and return mailed questionnaires.

#### 7.2 EARLY TERMINATION

Subjects may withdraw from the study voluntarily. In addition, if the PI determines that continued participation might present a safety risk for the subject then the PI may withdraw the subject from the study. Those subjects who receive study drug will be followed for 28 days after stopping study participation. Every effort will be made to obtain all end of treatment measures as outlined in (Table 1.Visit 6) in the event that a subject withdraws, or is withdrawn, from the study before completing treatment.

#### 8. STUDY PROCEDURES/EVALUATIONS


Compound No.: GTx-024

Please see Table1 Schedule of Measures for an outline of the timing of the study procedures. Please see Appendix A, B, C, D, E for outcomes measures.

#### **Interview with Vital Signs**

All potential subjects will be interviewed/assessed to confirm inclusion/absence of exclusion criteria. A review of systems will be completed, concomitant medications will be assessed, and vital signs (temperature, blood pressure, pulse and respirations) will be assessed. Laboratory results will also be reviewed at specified time points as outlined in Table 1.

#### **History**

A detailed history will include review of gravida, prior abortions,, parity, deliveries, and history of gynecological conditions and/or cancer.

#### **Focused Physical Exam**

A standard brief physical exam will be done. This will include a gynecological pelvic exam and visual skin exam with specific attention to androgenic changes.

#### **Urinalysis**

A clean catch midstream voided urine specimen will be obtained, and evaluated by urine dipstick. If results or clinical symptoms indicate, the specimen will be sent for culture and the patient will receive appropriate treatment for UTI per standard of care.

#### 24 Hour Pad Weight Test

The 24-hour pad test should be completed during 1 day of each scheduled 3-day diary. Subjects will be instructed to record pad weight on a day that is typical for them in terms of activity level and fluid intake. Subjects should be given one type of incontinence pad at the clinic. They may choose from a "light" pad or a "heavy" pad, but the pads dispensed **MUST** be used for the 24- hour test. Subjects should receive 8 incontinence pads for use during each 24-hour test period.

#### **Urethral Pressure Profile (UPP) and Bladder Stress Test**

To conduct the UPP and Bladder Stress Test, a urodynamic catheter will be placed and the bladder will be filled with 300 ml of fluid, such as saline. UPP will be performed. Subjects will be instructed to perform a provocative maneuver to increase abdominal pressure (cough, Valsalva, or similar event). Urine loss during this even indicates a positive stress test.

#### **Ultrasound Bladder Scan**

Subjects will be asked to void, and the volume of urine remaining in the bladder after voiding (post void residual) will be measured via bladder ultrasound scan.

Compound No.: GTx-024

#### Mammogram

Mammography is the process of using low-energy X-rays to examine the human breast, which is used as a diagnostic and screening tool. The goal of mammography is the early detection of breast cancer, typically through detection of characteristic masses and/or microcalcifications.

#### Magnetic Resonance Imaging(MRI)

MRI will be done at baseline and end of treatment to observe changes in pelvic floor muscles along with the thickness of the endometrium (mm). Quantiative assessments may include the area of the levator, the anteroposterior and transverse diameters, and/or other relevant parameters. Endometrial thickness can accurately be assessed by MRI (Stanislavsky, Weerakkody, et al., 2015; Nakamura et al., 2014); therefore, it is being used as a safety assessment in this study.

Medical, Epidemiological and Social Aspects of Aging (MESA) Questionnaire
The MESA questionnaire measures severity of specific types (stress, urgency, mixed) of
urinary incontinence (UI). Two subscales, the urgency UI (6 items) and the stress UI (9
items). Test-retest reliability on "any incontinence" is high (agreement coefficient = .89).
Validity (agreement between self-report on the MESA and clinician's assessment) =

Validity (agreement between self-report on the MESA and clinician's assessment) = 87% in women. The MESA questionnaire has demonstrated agreement on incontinence = 79% and 69% and 72% accuracy in predicting urodynamic diagnosis of stress UI and uninhibited detrusor contraction (Herzog, 1990a; Herzog, 1990b).

#### 3 Day Voiding Diary

Subjects will record each episode of urinary leakage and record its severity. Subjects will also be asked to record urinary frequency, and urgency. Urine volume will also be recorded. 3 day bladder diaries are reliable measures of mean number of UI episodes/day, UI type, mean voids/24 hours, and mean voids during sleeping hours. 2-week test-retest results correlate with diurnal micturition (r=.89, p<0.001) and UI episodes (r=.91, p<0.001). Compared to participant recall of the previous week, Spearman rank correlation = .57 for voiding frequency and .70 for UI episodes (Brown, 2003: Locher, 2001; Wyman, 1988). For this study, any episode of vaginal discharge or spotting will also be recorded on the diary.

#### Patient Global Impression of Improvement (PGI-I)

PGI-I is a global rating of improvement using 7-point scale. Construct validity was established in two randomized controlled studies (n=1,133 subjects) of drug treatment for predominant stress incontinence (Wagner, 1996; Yalcin, 2003).

#### Patient Global Impression of Severity (PGI-S)

PGI-S is a global rating of symptoms severity using a 7 point scale (Yalcin, 2003).

#### UDI-6 and IIQ-7

The Urogenital Distress Inventory (UDI-6) and Incontinence Impact Questionnaire (IIQ-7) assess symptom distress and the impact of urinary incontinence on daily life. The

Compound No.: GTx-024

urogenital distress inventory (UDI) and incontinence impact questionnaire (IIQ) were both developed to assess the impact of UI on HRQoL (Shumaker, 1994; Wyman, 1987). Short versions of the UDI and IIQ, UDI- 6, and IIQ-7, were developed to reduce the respondents' burden. The UDI-6 and IIQ-7 are both "A grade" recommended by the Fourth International Consultation on Incontinence (Shumaker, 1994; Wyman, 1987; Uebersax, 1995; Staskin, 2008).

#### Female Sexual Function Index (FSFI)

The FSFI is a 19-question validated tool evaluating sexual function in several domains: libido, arousal, lubrication, orgasm, satisfaction and pain (Rosen et al, 2000). Each subdomain is scored separately and the total score is calculated.

#### 9. ASSESSMENT OF SAFETY

## 9.1 METHODS AND TIMING FOR ASSESSING, RECORDING, AND ANALYZING SAFETY PARAMETERS

#### 9.1.1 ADVERSE EVENTS

ICH E6 defines an AE as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product regardless of its causal relationship to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.

The occurrence of an AE may come to the attention of study personnel during study visits and interviews of a study subject presenting for medical care, or upon review by a study monitor.

The period of observation for which AEs are to be collected begins after the subject has signed the ICF, throughout the study intervention period, and for 28 days post treatment.

All AEs, whether reported by the subject or noted by study personnel, will be recorded in the subject's medical record and captured on the appropriate CRF.

Information to be collected includes event description, time of onset, Investigator's assessment of severity, Investigator's assessment of relationship to study drug, and time of resolution/stabilization of the event. All AEs occurring while on study must be documented appropriately regardless of relationship to study drug. All AEs will be followed to adequate resolution as per Section 9.3 TYPE AND DURATION OF FOLLOW-UP OF SUBJECTS AFTER ADVERSE EVENTS.


Compound No.: GTx-024

Any medical condition that is present at the time that the subject is screened will be considered as baseline and not reported as an AE. However, if the condition deteriorates at any time during the study, it will be recorded as an AE. All AEs must be graded for intensity and relationship to study drug.

#### 9.1.2 INTENSITY OF EVENT

All AEs will be assessed by the Investigator according to NCI-CTCAE, Version 4.0. For any AE that is not specifically covered in NCI-CTCAE, Version 4.0, the criteria from

Table 1 should be used:

| Table 1: | Table 1: Description of Grades According to the CTCAE |
|---|---|
| Grade | Description |
| 0 | No AE or within normal limits |
| 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate; minimal, local, or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living |
| 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living |
| 4 | Life threatening consequences; urgent intervention indicated |
| 5 | Death related to AE |

If the intensity changes within a day, the maximum intensity should be recorded. If the intensity changes over a longer period of time, the changes should be recorded as separate events (having separate onset and stop dates for each change in intensity). Changes in the intensity of an AE will be documented to allow an assessment of the duration of the event at each level of intensity to be performed. AEs characterized as intermittent require documentation of onset and duration of each episode.

#### 9.1.3 DRUG – ADVERSE EVENT RELATIONSHIP

Classification of Relationship/Causality of Adverse Events (AE/SAE) to study drug: The investigator will determine the relationship between the study drug administration and the occurrence of an AE/SAE as defined below:

Not Related: The temporal relationship of the adverse event is determined to be Not Related to study drug administration.

Possibly Related: The temporal relationship of the adverse event to study drug administration makes a causal relationship possible. Other medications, therapeutic interventions, or underlying conditions provide a probable explanation for the observed event.

Compound No.: GTx-024

Probably Related: The temporal relationship of the adverse event to study drug administration makes a causal relationship.

Probable: Other medications, therapeutic interventions or underlying conditions provide a possible explanation for the observed event.

Related: The temporal relationship of the adverse event is determined to be Related to study drug administration.

Unable to Determine: The temporal relationship of the adverse event to study drug administration makes a causal relationship unable to determine or unknown.

#### 9.1.4 SERIOUS ADVERSE EVENTS

An SAE is defined as an AE that meets one of the following conditions:

- Death
- Life-threatening event (defined as a subject at immediate risk of death at the time of the event)
- An event requiring inpatient hospitalization or prolongation of existing hospitalization
- Results in congenital anomaly or birth defect
- Results in a persistent or significant disability/incapacity
- Any other important medical event that may not result in death, be life threatening, or require hospitalization, may be considered a serious adverse experience when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

#### All SAEs will be:

- Recorded on the appropriate CRF
- Reported to the designated Safety department/pharmacovigilance contractor using a SAE Report Form within 24 hours of awareness
- Followed through to resolution by a study Investigator
- Reviewed and evaluated by a study Investigator

Compound No.: GTx-024

#### 9.2 REPORTING PROCEDURES

#### 9.2.1 SERIOUS ADVERSE EVENTS

All SAEs, including death due to any cause, which occur after the subject signs the ICF and within 28 days following the last administration of study drug, whether or not related to the study drug, must be reported immediately to the designated Safety Department/pharmacovigilance contractor within **24 hours** by e-fax, e-mail, or telephone (see contact information below). At the very least, the following information must be reported:

- Date and time of report
- Reporter's name and phone number
- Investigator's name and site number
- Subject number
- SAE information: event term, onset date, causal relationship
- Study drug: start date of study drug and whether or not study drug has been withheld or discontinued

#### **SAE Reporting Contact Information:**

US Safety Toll-Free E-Fax Line: 1 866 966 2970

US Safety Toll-Free Unmanned Hotline: 1 866 966 8429

Safety E-mail: sae@cmedresearch.com

Information about all SAEs is collected and recorded on the SAE Report Form. The Investigator must assess the relationship of any SAE to study drug, complete the SAE Report Form, and send the completed, signed form by e-fax or e-mail within 24 hours to the assigned drug safety group. As a back-up, the site may report SAEs using the unmanned safety hotline, with a completed SAE Report Form forwarded to the assigned drug safety group within 24 hours following notification on the hotline. The original copy of the SAE Report Form and the e-fax confirmation sheet must be kept with the case report form documentation at the study site.

Follow-up information must also be sent to the same assigned drug safety group by e-fax or e-mail using either a new SAE Report Form stating that this is a follow-up to the previously reported SAE (giving the date of the original report), or by using a follow-up query form.

If an SAE is not previously documented (new occurrence) in the Investigator's Brochure (IB) and is thought to be related to the relevant Investigational Medicinal Product (IMP), the assigned drug safety group may urgently require further information from the Investigator for Regulatory Authority reporting. The drug safety group may need to issue an Investigator Notification (IN) to inform all Investigators involved in any study with the same drug that this SAE has been reported. Suspected Unexpected Serious Adverse Reactions (SUSARs) will be collected and reported to the regulatory/competent

Compound No.: GTx-024

authorities and relevant IRBs/IECs in accordance with Food and Drug Administration (FDA) regulations 21 CFR 312.32, International Conference on Harmonization (ICH) guidelines, and European Clinical Trials Directive 2001/20/EC, or as per national regulatory requirements in participating countries. Adequate documentation must be maintained showing that Regulatory Authorities and IRBs/IECs have been properly notified.

**SAEs must be reported within 24 hours**, regardless of relationship, on a SAE Report Form to allow the Sponsor to take appropriate measures to address potential new risks in a clinical trial. The Investigator must report such events to the Sponsor immediately; under no circumstances should reporting take place more than 24 hours after the Investigator learns of the event.

The term sudden death should be used only when the cause is of a cardiac origin as per standard definition. The terms death and sudden death are clearly distinct and must not be used interchangeably. The study will comply with all local regulatory requirements and adhere to the full requirements of the ICH Guideline for Clinical Safety Data Management, Definitions and Standards for Expedited Reporting, Topic E2.

The SAE Report Form must be signed by the PI or assigned designee.

Other supporting documentation of the event may be requested by the safety department/pharmacovigilance contractor and should be provided as soon as possible.

All SAEs will be followed until satisfactory resolution as per Section 9.3 TYPE AND DURATION OF FOLLOW-UP OF SUBJECTS AFTER ADVERSE EVENTS.

#### 9.2.2 REGULATORY REPORTING

Suspected (considered related to the study drug) and unexpected (not previously described in the reference safety document) serious adverse reactions (SUSARs) will be reported in an expedited manner by GTx, Inc. to applicable Regulatory Authorities, EudraVigilance, IECs and IRBs, and Investigators in compliance with FDA regulations 21 CFR 312.32, ICH guidelines, the European Clinical Trials Directive 2001/20/EC, the European Commission's "Detailed guidance on the collection, verification and presentation of adverse event/reaction reports arising from clinical trials on medicinal products for human use" (CT-3, June 2011), and other applicable local regulations and guidelines, as required. The timelines stipulated by applicable national regulations and guidelines shall be adhered to, typically death and life-threatening SUSARs shall be reported within 7 days and all other SUSARs shall be reported within 15 days.

Additionally, events may occur during a clinical trial which do not fall within the definition of a SUSAR and thus are not subject to the reporting requirements for SUSARs, even though they may be relevant in terms of subject safety. Examples are new events

Compound No.: GTx-024

related to the conduct of a trial or the development of an IMP likely to affect the safety of subjects such as:

- A SAE which could be associated with the trial procedures and which could modify the conduct of the trial
- A significant hazard to the subject population such as lack of efficacy of an IMP used for the treatment of a life-threatening disease
- A major safety finding from a newly completed animal study (such as carcinogenicity)

These events/observations are not to be reported as SUSARs, but they might require other action, such as urgent safety measures and their notification, substantial amendments, or early termination of the trial, and shall be reported in accordance with applicable local regulations and guidelines.

All serious events designated as expected and/or "not related" to study drug(s), will be reported to the applicable Regulatory Authorities and IECs/IRBs at least annually in a summary format".

## 9.3 TYPE AND DURATION OF FOLLOW-UP OF SUBJECTS AFTER ADVERSE EVENTS

AEs will be collected up until 28 days after the last dose of study treatment, and will continue to be followed up until one of the following occurs:

Resolved or improved to baseline Death

Investigator confirms that no further improvement can be expected

#### 9.4 HALTING RULES

If in the opinion of the Investigator, the participation in the study is or is becoming detrimental to the well-being of a particular subject, this issue should be discussed with the Medical Monitor for this study and the subject's participation in the study may be discontinued.

Discontinuation of treatment should be considered if:

ALT or AST > 8 × ULN

ALT or AST > 5 × ULN for more than 2 weeks

ALT or AST  $> 3 \times ULN$  and ((total bilirubin  $> 2 \times ULN$  or INR > 1.5)

ALT or AST >  $3 \times ULN$  with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%)


Compound No.: GTx-024

All subjects discontinued from the study should be followed until abnormal values return to normal.

ALL DISCONTINUATIONS SHOULD BE DISCUSSED WITH THE MEDICAL MONITOR PRIOR TO DISCONTINUATION.

#### 10. STATISTICAL CONSIDERATIONS

Since this is a proof of concept feasibility study, no power calculation is needed. Based on Dalton, 2011, 10-20% of patients may withdraw from the study before completing treatment. Therefore, we will recruit up to 35 patients meeting inclusion/exclusion criteria until 30 subjects have completed treatment. Descriptive statistics will be used to explore changes in primary and secondary outcomes measures between baseline and end of treatment. Although the primary efficacy measure will be a change in frequency of daily stress leaks between Baseline and Week 14 weeks, response to treatment will also consider secondary efficacy measures (change in frequency of voids per day, urine volume per void, change in 24 hour pad weight, responses to validated questionnaires, changes in UPP measures, changes in sexual function), and change in pelvic floor muscles as measured by MRI. Safety will be reported by the number and type of adverse events reported during treatment. No imputations for missing data will be conducted. There will be no adjustment for multiple testing.

#### 10.1 STATISTICAL METHODS

#### Primary end point

 The average number of episodes per day of leaking (SUI) will be calculated by summing the number of episodes over the 3 day period and dividing by 3, the change from Baseline to Week 12 will be computed and this change will be summarized with descriptive statistics (min, max, median, mean, standard deviation) and analyzed for a significant change from Baseline using the Exact Wilcoxon sign rank test.

#### Secondary end points

- The average number of voids per day will be calculated by summing the number
  of voids over the 3 day period and dividing by 3, the change from Baseline to
  Week 12 will be computed and this change will be summarized with descriptive
  statistics (min, max, median, mean, standard deviation) and analyzed for a
  significant change from Baseline using the Exact Wilcoxon sign rank test.
- The average volume per void will be calculated by summing the total urine amount over the 3 day period and dividing by the total number of voids recorded over 3 days, the change from Baseline to Week 1[2 will be computed and this


Compound No.: GTx-024

change will be summarized with descriptive statistics (min, max, median, mean, standard deviation) and analyzed for a significant change from Baseline using the Exact Wilcoxon sign rank test.

- Change in maximum urethral closure pressure measurements from Baseline to Week 12 will be computed and this change will be summarized with descriptive statistics (min, max, median, mean, standard deviation) and analyzed for a significant change from Baseline using the Exact Wilcoxon sign rank test.
- Change in 24 hour pad weight from Baseline to Week 12 will be computed and this change will be summarized with descriptive statistics (min, max, median, mean, standard deviation) and analyzed for a significant change from Baseline using the Exact Wilcoxon sign rank test.
- Change in total score on the stress incontinence section of the MESA Urinary
  Questionnaire from Baseline to Week 12 will be computed and this change will
  be summarized with descriptive statistics (min, max, median, mean, standard
  deviation) and analyzed for a significant change from Baseline using the Exact
  Wilcoxon sign rank test.
- Change in Patient Global Impression of Severity (PGI-S) Scale from Baseline to Week 12 will be computed and this change will be summarized with descriptive statistics (min, max, median, mean, standard deviation) and analyzed for a significant change from Baseline using the Exact Wilcoxon sign rank test
- Patient Global Impression of Improvement (PGI-I) Scale at Week 12. Descriptive statistics, (min, max, median, mean, standard deviation) will summarize these scores.
- Change in total score on the Urinary Distress Inventory (UDI-6) from Baseline to Week 12 will be computed and this change will be summarized with descriptive statistics (min, max, median, mean, standard deviation) and analyzed for a significant change from Baseline using the Exact Wilcoxon sign rank test.
- Change in total score on the Incontinence Impact Questionnaire (IIQ-7) from Baseline to Week 12 will be computed and this change will be summarized with descriptive statistics (min, max, median, mean, standard deviation) and analyzed for a significant change from Baseline using the Exact Wilcoxon sign rank test.
- Change in total score on the Female Sexual Function Index (FSFI) as well as the change in subdomain scores: libido, arousal, lubrication, orgasm, satisfaction, and pain from Baseline to Week 12 will be computed and these changes will be summarized with descriptive statistics (min, max, median, mean, standard deviation) and analyzed for a significant change from Baseline using the Exact Wilcoxon sign rank test.


Compound No.: GTx-024

- Changes in pelvic floor muscles from Baseline to Week 12 will be summarized with descriptive statistics (min, max, median, mean, standard deviation) and analyzed for a significant change from Baseline using the Exact Wilcoxon sign rank test.
- Qualitative changes in pelvic muscles will be described as decreased, increased or no change at Week 12 relative to Baseline.

#### **Exploratory Analyses**

Changes from baseline to each of the assessment times prior to Week 12 for the above endpoints will be explored, described and tested for significance using the same analytical methods noted for the primary and secondary objectives above. Durability treatment will be assessed by evaluating changes in study measures between week 12 and 16 (end of study). There will be no adjustment for multiple testing, nor will any data be imputed.

Repeated measures (mixed models) will be used to examine the change over time by incorporating all available assessment times to test for a significant non-zero slope over time and estimate that slope and its standard error.

Various imputation methods may be explored if any of the above analyses indicate promise for the compound in the treatment of SUI. These imputation methods may allow for better estimation of effect size and consequently sample size estimation in future trials.

#### 11. QUALITY CONTROL AND QUALITY ASSURANCE

Standard operating procedures are available for all activities relevant to the quality of this study. Designated personnel will be responsible for implementing and maintaining quality assurance and quality control systems to ensure that the study is conducted, and that data are generated, documented, and reported in compliance with the study protocol, GCP, and Good Laboratory Practice requirements as well as applicable regulatory requirements and local laws, rules, and regulations relating to the conduct of the clinical study.

An authorized Quality Assurance auditor will audit the study data and procedures at periodic intervals as indicated. Domestic or foreign regulatory authorities, the IRB/IEC, and a Sponsor-authorized auditor may request access to all study documentation for an on-site inspection or audit. The Investigator must notify GTx, Inc. of any regulatory authority inspections and forward copies of the inspection report to GTx, Inc.

Compound No.: GTx-024

Electronic data systems will be in accordance with applicable aspects of 21 CFR Part 11, ICH Guidelines, GCP, local laws and legislation, and the Health Insurance Portability and Accountability Act.

#### **On-site Audits**

At any time, quality assurance representatives of the Sponsor and/or regulatory bodies may visit the unit to carry out an audit of the study in compliance with regulatory guidelines and company policy. Such audits will require access to study records, documentation, and regulatory files. At all times, subject privacy will be of utmost importance and respected. Typically, sufficient notice will be given to the Investigator to prepare for the visit.

#### 12. ETHICS/PROTECTION OF HUMAN SUBJECTS

#### 12.1 ETHICAL CONSIDERATIONS

This clinical study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki and in accordance with global regulations including 21 CFR 312.

The investigator is responsible for obtaining approval for this clinical study from the relevant IRB at the associated institution. The study will not begin until a favorable opinion of the IRB has been obtained. The investigator is responsible for complying with requirements imposed by the IRB and/or regulatory authority. Furthermore, the investigator will ensure that local regulations concerning data protection are followed. For ethical considerations, all patients will be required to sign a consent indicating their willingness to participate and that they have been fully informed of the risks and benefits of participation.

## 12.2 INSTITUTIONAL REVIEW BOARD/ INDEPENDENT ETHICS COMMITTEE

The protocol and the proposed ICF will be reviewed and approved by a properly constituted IRB/IEC before the study start. A signed and dated statement that the protocol and informed consent have been approved by the IRB/IEC will be given to GTx, Inc. or designee before study initiation. The signed IRB/IEC approval letter must identify the documents approved (i.e., list the Investigator's name, the protocol number and title, the date of the protocol, and the date of approval of the protocol and the informed consent document). Any advertisements used to recruit subjects must also be reviewed by the IRB/IEC. Clinical supplies will not be shipped to a site until a signed approval letter from the IRB/IEC has been received and a contractual agreement has been signed by both parties.

Compound No.: GTx-024

Prior to study start, the Investigator will be required to sign a protocol signature page confirming his/her agreement to conduct the study in accordance with these documents and all of the instructions and procedures found in this protocol and to give access to all relevant data and records to GTx, Inc. monitors, auditors, GTx, Inc. Clinical Quality Assurance representatives, designated agents of GTx, Inc., IRBs/IECs/Research Ethics Boards (REBs), and regulatory authorities as required.

#### 12.3 PRE-STUDY DOCUMENTATION

The Investigator must provide GTx or its designee with the following documents prior to the enrollment of any subjects:

- Copy of the signed Investigator Agreement page
- Copy of the IRB/IEC approval letter for protocol and informed consent
- Completed, signed, and dated Form FDA 1572
- Current curricula vitae, licenses, and financial disclosures for the Investigator(s) and sub Investigators listed on the 1572
- Where applicable, list of IRB/IEC committee members and a statement of adherence to GCP
- Copy of approved informed consent document
- Executed clinical trial agreement
- Name, location, certification number, and date of certification of the laboratory to be used for laboratory assays and those of other facilities conducting tests. GTx or its designee must be notified if the central laboratory is changed or if any additional laboratory is to be used
- List of normal laboratory values (i.e., reference ranges and units of measure) for each central laboratory to be used during the study. GTx or its designee must be notified if normal values change

#### 12.4 INFORMED CONSENT PROCESS

Eligible subjects will only be included in the study after providing written (witnessed, where required by law or regulation), IRB/IEC-approved informed consent.

The informed consent documents must be reviewed and approved by GTx or its designee and the investigative site IRB/IEC prior to the initiation of the study.

Each subject will receive an IRB/IEC approved informed consent document with study information. Subjects should be given ample time to read the information and the opportunity to ask questions. Informed consent must be obtained from each subject prior to performing any protocol-specific evaluations. The signed ICF will be retained with the study records and the subject will receive a copy of the signed informed consent for his/her records. The process of obtaining informed consent will be documented in the subject source documents.

Compound No.: GTx-024

The date when a subject's informed consent was actually obtained will be captured in their CRFs.

The Investigator (or designated staff) will explain the nature of the study as well as its risks and benefits to the subject (or the subject's legal representative).

#### 12.5 SUBJECT CONFIDENTIALITY

Subject confidentiality is strictly held in trust by the participating Investigators, their staff, and the Sponsor(s) and their agents. This confidentiality is extended to cover testing of biological samples and genetic tests (if applicable) in addition to the clinical information relating to participating subjects.

The study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the Sponsor.

The study monitor or other authorized representatives of the Sponsor may inspect all documents and records required to be maintained by the Investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the subjects in this study. The clinical study site will permit access to such records.

#### 12.6 PROTOCOL ADHERENCE

By signing the Form FDA 1572, the Investigator agrees to conduct the study according to the protocol and the FDA regulations set forth in 21 CFR Parts 50, 54, 56, and 312.

#### 12.7 PERMISSION TO REVIEW SUBJECTS' SOURCE RECORDS

The Investigator agrees to allow the FDA and other regulatory agencies, individuals delegated by the IRB/IEC and Competent Authorities, and the Sponsor or its designee to have access to all the original documentation of the study, including the ICFs signed by the subjects enrolled into the study and the relevant subject medical files. The individuals who are given access to the documentation must take every reasonable precaution to keep the identity of the subjects and the proprietary information of the Sponsor as confidential information in accordance with relevant applicable legislation.

#### 12.8 PROTOCOL AMENDMENTS

All amendments to the study protocol must be submitted to the IRB/IEC for written approval. The approval letter, signed by the IRB/IEC Chairperson, must refer specifically to the Investigator, the protocol number and protocol title, the protocol

Compound No.: GTx-024

amendment number, and the date of the protocol amendment. A copy of the approval letter and revised informed consent document (if applicable) must be sent to GTx or its designee. A protocol amendment may be implemented only after it has been approved by the IRB/IEC and has been approved by the appropriate regulatory authority. In the case of a protocol change intended to eliminate an apparent immediate hazard to subjects, the change may be implemented immediately, but the change must then be documented in a protocol amendment and approved as described above.

#### 12.9 CHANGE IN INVESTIGATOR

If any Investigator retires, relocates, or withdraws from an investigation during the conduct of the study the responsibility for conduct of the study may be transferred to another appropriately qualified Investigator at the investigative site. GTx or its designee must be notified. An updated Form FDA 1572 must be submitted to GTx or its designee.

#### 12.10 STUDY DISCONTINUATION

GTx, Inc. reserves the right to discontinue this study under the conditions specified in the clinical study agreement.

#### 12.11 INDEMNITY

The Sponsor certifies that it has taken out a liability insurance policy that is consistent with the requirements for which the study is being conducted. This insurance policy is in accordance with local laws and requirements. An insurance certificate will be provided to the PI requiring this document. The insurance of the Sponsor does not relieve the PI and the collaborators of any obligation to maintain their own liability insurance policy as required by applicable law.

#### 13. DATA HANDLING AND RECORD KEEPING

The Investigator is responsible to ensure the accuracy, completeness, legibility, and timeliness of the source data. All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data. Dark ink is required to ensure clarity of reproduced copies. When making changes or corrections, cross out the original entry with a single line, and initial and date the change. DO NOT ERASE, OVERWRITE, OR USE CORRECTION FLUID OR TAPE ON THE ORIGINAL.

Copies of the CRF will be provided for use as source documents and maintained for recording data for each subject enrolled in the study. Data reported in the CRF derived from source documents should be consistent with the source documents or the discrepancies should be explained.

Compound No.: GTx-024

Study records will be maintained in locked offices with access limited to authorized individuals. Each participant will be given an identification number that will be used to enter the data into a password protected database and for the analysis.

#### 13.1 DATA CAPTURE METHODS

#### 13.1.1 DATA COLLECTION

Study specific data will be collected on paper case report forms (CRFs). Completed questionnaires and voiding diaries will be used as source documents, and these documents will be kept in the study files. Blank data fields should be noted as unknown (UNK) or not applicable (NA) if source information is not available or data not collected. While completing the questionnaire, if a subject leaves a question blank, it will be deemed permanently missing. All CRFs will be maintained at the study site for the length of time as determined by the IRB and federal regulations and as provided in the site's clinical study agreement. Data will be entered into a password protected electronic database that does not contain subject identifiers. Identifiers linked to unique Study ID will be kept separately from the study data. Data entry will be reviewed for accuracy.

#### 13.2 STUDY SITE RESPONSIBILITIES

All data requested on the CRF must be recorded. Data will be transcribed by authorized personnel at the study site from the source documents into the CRF for enrolled subjects. All information on the CRF must be traceable to these source documents. All electronic entries (including any changes or updates) will be traceable through the system. Only the PI or authorized staff may enter or modify data in the database using their unique password. The Investigator must certify that the data entered in the CRFs are complete and accurate by electronically signing the CRF.

#### 13.3 CRF TIMING/REPORTS

A final report for the study will be completed upon completion of the study and the analysis of data. Please see information concerning publication policy (Section 14).

#### 13.4 STUDY RECORDS RETENTION

Study documents must be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period, however, if required by local regulations. No records will be destroyed without the written consent of GTx, Inc., if applicable. It is the responsibility of GTx, Inc. to inform the PI when these documents no longer need to be retained.

Compound No.: GTx-024

#### 13.5 PROTOCOL DEVIATIONS

A protocol deviation is any noncompliance with the clinical trial protocol that affects a subject's safety and primary efficacy, GCP, or Manual of Procedures requirements. The noncompliance may be either on the part of the subject, the PI, or the study site staff. As a result of deviations, corrective actions are to be developed by the site and implemented promptly.

These practices are consistent with ICH E6:

- 4.5 Compliance with Protocol, sections 4.5.1, 4.5.2, and 4.5.3
- 5.1 Quality Assurance and Quality Control, section 5.1.1
- 5.20 Noncompliance, sections 5.20.1 and 5.20.2

It is the responsibility of the site to use continuous vigilance to identify and report deviations within 5 working days of identification of the protocol deviation. All deviations from the protocol must be addressed in study subject source documents. A completed copy of the Protocol Deviation Form will be maintained in the regulatory file, as well as in the subject's source document. Protocol deviations will be sent to the local IRB/IEC per their guidelines. The PI/study staff is responsible for knowing and adhering to their IRB/IEC requirements.

Compound No.: GTx-024

#### 14. PUBLICATION POLICY

Following completion of the study, it is expected some Investigators may wish to publish the results of this research in scientific journal(s). Publication rights are governed by the investigatory site's clinical trial agreement with GTx, Inc. The Investigator may request to publish this study in a scientific journal, but must have written authorization of GTx, Inc.

The data generated by this study are confidential information and the property of GTx, Inc. This confidential information may be published only in collaboration with participating personnel from GTx, Inc. or upon GTx's written consent, or otherwise under terms of the investigatory site's clinical trial agreement with GTx, Inc. All unpublished information shall not be disclosed to any third parties without the prior written consent of GTx, Inc.

The International Committee of Medical Journal Editors member journals have adopted a trials-registration policy as a condition for publication. This policy requires that all clinical trials be registered in a public trials registry such as *ClinicalTrials.gov*, which is sponsored by the U.S. National Library of Medicine. It is GTx's responsibility to register this trial in an acceptable registry.


Compound No.: GTx-024

#### 15. LITERATURE REFERENCES

Aizawa K, Iemitsu M, Maeda S, Mesaki N, Ushida T, Akimoto T. Endurance exercise training enhances local sex steroidogenesis in skeletal muscle. Medicine and science in sports and exercise 2011; 43(11): 2072-80.

Antonio FI, Bo K, Ferriani RA, de Sa MF, de Sa Rosa e Silva AC, Ferreira CH. Pelvic floor muscle strength and urinary incontinence in hyperandrogenic women with polycystic ovary syndrome. International urogynecology journal 2013; 24(10): 1709-14.

Athanasiou S, Khullar V, Boos K, Salvatore S, Cardozo L. Imaging the urethral sphincter with three-dimensional ultrasound. Obstet Gynecol 1999; 94(2): 295-301

Bai SW, Jung BH, Chung BS, et al. Relationship between urinary profile of the endogenous steroids and postmenopausal women with stress urinary incontinence. Neurourol Urodynam 2003; 22: 198-205.

Bai SW, Jung BH, Chung BC, et al. Relationship between urinary endogenous steroid metabolites and lower urinary tract function in postmenopausal women. Yonsei Med J 2003; 44: 279-87.

Berger L, El-Alfy M, Martel C, Labrie F. Effects of dehydroepiandrosterone, Premarin and Acolbifene on histomorphology and sex steroid receptors in the rat vagina. J Steroid Biochem Mol Biol. 2005; 96: 201-15.

Berman JR, Almeida FG, Jolin J, et al. Correlation of androgen receptors, aromatase, and 5-alpha reductase in the human vagina with menopausal status. Fertil Steril 2003; 79: 925–931.

Brown JS, McNaughton KS, Wyman JF, Burgio KL, Harkaway R, Bergner D, Altman DS. Kaufman J, Kaufman K, and Girman CJ, Measurement characteristics of a voiding diary for use by men and women with overactive bladder. Urology, 2003. 61(4): 802-9.

Brubaker L, Norton PA, Albo ME, Chai TC, Dandreo KJ. Adverse events over two years after retropubic or transobturator midurethral sling surgery: findings from the Trial of Midurethral Slings (TOMUS) study. Am J Obstet Gynecol 2011, 205: 498.e1–498.e6

Cammu H, Van Nylen M, Blockeel C, Kaufman L, Amy J-J. Who will benefit from pelvic floor muscle training for stress urinary incontinence? Am J Obstet Gynecol 2004; 191: 1152-7.

Celayir S, Ilce Z, Dervisoglu S. The sex hormone receptors in the bladder in childhood-I: preliminary report in male subjects. Eur J Pediatr Surg 2002; 12: 312–317.

Compound No.: GTx-024

Copas P, Bukovsky A, Asbury B, et al. Estrogen, progesterone, and androgen receptor expression in levator ani muscle and fascia. J Women Health Gend Based Med 2001; 10: 785–795.

Dalton JT, Barnette KG, Bohl CE, et al. The selective androgen receptor modulator GTx-024 improves lean body mas and physical function in healthy elderly men and postmenopausal women: results of a double-blind, placebo-controlled phase II trial. J Cachexia Sarcopenia Muscle 2011; 2: 153-61.

DeLancey JO, Miller JM, Kearney R, Howard D, ReddyP, Umek W, Guire KE, Margulies RU, Ashton-Miller JA. Vaginal birth and de novo stress incontinence: relative contributions of uretliral dysfiinction and mobility. Obstet Gynecol 2007; (2Pt I); 354~362.

DeLancey JO, Trowbridge ER, Miller JM, Morgan DM, Guire K, Fenner DE, Weadock WJ, Ashton-Miller JA. Stress urinary incontinence: relative importance of urethral support and urethral closure pressure. J Urol. 2008; 179 (6); 2286-2290.

Dmochowski RR, Miklos JR, Norton PA, et al. for the Duloxetine Urinary Incontinence Study Group. Duloxetine versus placebo for the treatment of North American women with stress urinary incontinence. J Urol 2003; 170: 1259-1263.

Hay-Smith J, Berghmans B, Burgio K, Dumoulin C, Hagen S, Moore K, Nygaard I, N'dow J (2009) Committee 12 adult conservative management. In: Abrams P, Cardozo L, Khoury S, Wein A (eds) Incontinence, 4th edn. Health Publications Ltd., Paris

Herzog AR, Diokno AC, Brown MB, Normolle DP, and Brock BM, Two-year incidence, remission, and change patterns of urinary incontinence in noninstitutionalized older adults. J Gerontol 1990, 34: M67-74.

Herzog AR, Fultz NH. Prevalence and incidence of urinary incontinence in community-dwelling populations. J Am Geriatr Soc, 1990. 38(3): p. 273-81. PMID 2179368 adults. J Gerontol, 1990. 45(2): M67-74.

Ho MH, Bhatia NN, Bhasin S. Anabolic effects of androgens on muscles of female pelvic floor and lower urinary tract. Current opinion in obstetrics & gynecology 2004; 16(5): 405-9.

Jung BH, Bai SW, Chung BC. Urinary profile of endogenous steroids in postmenopausal women with stress urinary incontinence. J Reprod Med 2001; 46: 969–974.

Kadekawa et al, AUA Annual Meeting 2015, New Orleans, LA. PD27-11.

Compound No.: GTx-024

Kenton K, Mueller E, Bmbaker L. Continent women have better urethral neuromuscular function than those with stress incon¬tinence. Int Urogynecol J. 2011; 22(12): 1479-1484.

Kvarstein B.K., Nygaard I. Lower urinary tract symptoms and pelvic floor muscle exercise adherence after 15 years. Obstet Gynecol 2005; 105: 999-1005

Labrie J, Berghmans BLCM, Fischer K, Milani A, van der Wijk I, et al. Surgery versus physiotherapy for stress urinary incontinence. NEJM 2013; 369: 1124-1133.

Lamers BHC, van der Vaart CH. Medium- term efficacy of pelvic floor muscle training for female urinary incontinence in daily practice. Int Urogynecol J Pelvic Floor Dysfunct 2007; 18: 301-7.

Lee PE, Kumg RC, Drutz HP. Periurethral autologous fat injection as a treatment for female stress urinary incontinence-a randomized double-blind controlled trial. J Urol 2001; 165; 153-158

Locher JL, Goode PS, Roth DL, Worrell RL, and Burgio KL, Reliability assessment of the bladder diary for urinary incontinence in older women. J Gerontol A Biol Sci Med Sci, 2001. 56(1): M32-5.

Luber KM: The definition, prevalence, and risk factors for stress urinary incontinence. Rev Urol, suppl., 2004; 6: S3.

Madill SJ, Pontbriand-Drolet S, Tang A, Dumoulin C. Changes in urethral sphincter size following rehabilitation in older women with stress urinary incontinence. Int Urogynecol J 2014, September, epub ahead of print.

Mammadov R, Sinsir A, Tuglu I, Eyren V, Gurer E, Ozyurt C. The effect of testosterone treatment on urodynamic findings and histopathomorphology of pelvicjHoor muscles in female rats with experimentally induced stress urinary incontinence. Int Urol Nephrol 2011; 43: 1003-1008

McLean L, Varette K, Gentilcore-Saulnier B, Harvey MA, Baker K, Sauerbrei E (2013) Pelvic floor muscle training in women with stress urinary incontinence causes hypertrophy of the urethral sphincters and reduces bladder neck mobility during coughing. Neurourol Urodyn 32(8): 1096-n02. doi; 10.1002/nau.22343

Mohler ML, Bohl CE, Jones A, et al. Nonsteroidal selective androgen receptor modulators (SARMs): dissociating the anabolic and androgenic activities of the androgen receptor for therapeutic benefit. J Med Chem 2009; 52(12): 3597-617.

Compound No.: GTx-024

Montezuma T, Antonio FI, Rosa e Silva AC, Sa MF, Ferriani RA, Ferreira CH. Assessment of symptoms of urinary incontinence in women with polycystic ovary syndrome. Clinics (Sao Paulo, Brazil) 2011; 66(11): 1911-5.

Morgan DM, Umek W, Guire K, Morgan HK, Garabrant A, DeLancey JO. Urethral sphincter morphology and function with and without stress incontinence. J Urol. 2009; 182(I); 203-209.

Norton PA, Zinner NR, Yalcin I, Bump RC; Duloxetine Urinary Incontinence Study Group. Duloxetine versus placebo in the treatment of stress urinary incontinence. Am J Obstet Gynecol 2002, 187: 40-8

Nnodim JO. Quantitative study of the effects of denervation and castration on the levator ani muscle of the rat. Anat Rec 1999; 255: 324–333.

Nnodim JO. Testosterone mediates satellite cell activation in denervated rat levator ani muscle. Anat Rec 2001; 263: 19–24.

Peters KM, Dmochowski RR, Carr LK, Magali R, Kaufman MR, Sirls LT, Herschorn S, Birch C, Kultgen PL, Chancellor MB.Autologous muscle derived cells for treatment of stress urinary incontinence in women. J Urol 2014; 192: 469-476.

Rosen R, Brown C, Heiman J, Leiblum S, Meston CM, Shabisigh R, Ferguson D, D'Agostino R, Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Mar Ther 2000; 26, 191-208.

Rovner ES, Wein AJ. Treatment options for stress urinary incontinence. Reviews in Urology 2004; 6: s 29-s47

Santen RJ, Vaginal administration of estradiol: effects of dose, preparation and timing on plasma estradiol levels Climacteric 2015; 18:121-134

Shin MH, Rhie GE, Park CH, Kim KH, Cho KH, Eun HC, et al. Modulation of collagen metabolism by the topical application of dehydroepiandrosterone to human skin. J Invest Dermatol. 2005; 124: 315-23.

Shumaker SA, Wyman JF, Uebersax JS. et al. Health-related quality of life measures for women with urinary incontinence: The Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program in Women (CPW) Research Group. Qual Life Res 1994; 3: 291–306.

Staskin D, Kelleher C. Incontinence, Patient-Reported Outcome Assessment. 4th International Consultation on Incontinence; July 5–8, 2008, 2009; Paris Data Collection Tools/Case Report Forms

Compound No.: GTx-024

Takahashi S, Homnia Y, Fujishiro T, Hosaka Y, Kitamura T, Kawabe K. Electromyographic study of the striated urethral sphincter in type 3 stress incontinence: evidence of myogenic-dominant damages. Urology 2000, 56(6); 946-950

Uebersax JS, Wyman JF, Shumaker SA. et al. Short forms to assess life quality and symptom distress for urinary incontinence in women: The Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn 1995; 14: 131–9.

Wagner TH, Patrick DL, Bavendam TG, Martin ML, Buesching DP. Quality of life of persons with urinary incontinence: development of a new measure. Urology, 1996. 47(1): 67-71; discussion 71-2.

Wyman JF, Choi SC, Harkins SW, Wilson MS, and Fantl JA, The urinary diary in evaluation of incontinent women: a test-retest analysis. Obstet Gynecol, 1988. 71(6 Pt 1): 812-7.

Wyman JF, Harkins SW, Choi SC. et al. Psychosocial impact of urinary incontinence in women. Obstet Gynecol 1987; 70: 378–81.

Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol, 2003. 189(1): 98-101.

Protocol: GTx-024 as a Treatment for Stress Urinary
Incontinence in Women: A Proof of Concept Study

Compound No.: GTx-024
Author: \_\_\_\_\_

#### 1. APPENDIX A: MESA URINARY QUESTIONNAIRE

| MESA | Urinary Questionnaire | | | | |
|---|---|---|---|---|---|
| NAME | E (printed): | | | | |
| 1. | Over the past three months, have | you had urine loss beyond yo | our control? Yes No | | |
| 2. | How long ago did your urine loss | start? Years Months Da | ays | | |
| | Urge Incontinence | | | | |
| 1. | Some people receive very little wa | arning and suddenly find that | they are losing, or about to lose, urine | beyond their control. How often does this h | appen to you? |
| | Often | Sometimes | Rarely | Never | |
| 2. | If you can't find a toilet or find a to | ilet that is occupied and you h | have an urge to urinate, how often do | you end up losing urine and wetting yoursel | f? |
| | Often | Sometimes | Rarely | Never | |
| 3. | Do you lose urine when you sudde | enly have the feeling that you | r bladder is full? | | |
| | Often | Sometimes | Rarely | Never | |
| 4. | Does washing your hands cause y | ou to urinate? | | | |
| | Often | Sometimes | Rarely | Never | |
| <b>5</b> . | Does cold weather cause you to le | ose urine? | | | |
| | Often | Sometimes | Rarely | Never | |
| 6. | Does drinking cold beverages cau | se you to lose urine? | | | |
| | Often | Sometimes | Rarely | Never | |
| | Stress Incontinence | | | | |
| 1. | Does coughing gently cause you t | o lose urine? | | | |
| | Often | Sometimes | Rarely | Never | |
| 2. | Does coughing hard cause you to | lose urine? | | · | |
| | Often | Sometimes | Rarely | Never | |

Protocol: GTx-024 as a Treatment for Stress Urinary
Incontinence in Women: A Proof of Concept Study

Compound No.: GTx-024
Author: \_\_\_\_\_\_

| 3. | Does sneezing cause you to lose urine? | | | |
|---|---|---|---|---|
| | Often | Sometimes | Rarely | Never |
| 4. | Does lifting things cause you to lose | urine? | | |
| | Often | Sometimes | Rarely | Never |
| 5. | Does bending over cause you to lose | e urine? | | |
| | Often | Sometimes | Rarely | Never |
| 6. | Does laughing cause you to lose urine? | | | |
| | Often | Sometimes | Rarely | Never |
| 7. | Does walking briskly cause you to lose urine? | | | |
| | Often | Sometimes | Rarely | Never |
| 8. | Does straining, if you are constipated, cause you to lose urine? | | | |
| | Often | Sometimes | Rarely | Never |
| 9. | Does getting up from a sitting to a standing position cause you to lose urine? | | | |
| | Often | Sometimes | Rarely | Never |

| Protocol: GTx-024 as a Treatment for Stress Urinary Incontinence in Women: A Proof of Concept Study | Compound No.: GTx-024<br>Author: |
|---|---|
|---|---|

#### Total Calculator:

| URGE SYMTOM INDEX LO | URGE SYMTOM INDEX LOOK-UP TABLE | | | |
|---|---|---|---|---|
| 1/18 = 6% | 5/18 = 28% | 9/18 = 50% | 13/18 = 72% | 17/18 = 94% |
| 2/18 = 11% | 6/18 = 33% | 10/18 = 56% | 14/18 = 78% | 18/18 = 100% |
| 3/18 = 17% | 7/18 = 39% | 11/18 = 61% | 15/18 = 83% | |
| 4/18 = 22% | 8/18 = 44% | 12/18 = 67% | 16/18 = 89% | |

Total Score \_\_\_\_\_/18

| STRESS SYM | STRESS SYMPTOM INDEX LOOK-UP TABLE | | | | | |
|---|---|---|---|---|---|---|
| 1/27 = 4% | 5/27 = 19% | 9/27 = 33% | 13/27 = 48% | 17/27 = 63% | 21/27 = 78% | 25/27 = 93% |
| 2/27 = 7% | 6/27 = 22% | 10/27 = 37% | 14/27 = 52% | 18/27 = 67% | 22/27 = 81% | 26/27 = 96% |
| 3/27 = 11% | 7/27 = 26% | 11/27 = 41% | 15/27 = 56% | 19/27 = 70% | 23/27 = 85% | 27/27 = 100% |
| 4/27 = 15% | 8/27 = 30% | 12/27 = 44% | 16/27 = 59% | 20/27 = 74% | 24/27 = 89% | |

Total Score \_\_\_\_\_/27

Protocol: GTx-024 as a Treatment for Stress Urinary
Incontinence in Women: A Proof of Concept Study

Compound No.: GTx-024
Author: \_\_\_\_\_\_

# 2. APPENDIX B: PATIENT GLOBAL IMPRESSION OF SEVERITY (PGI-S) SCALE AND PATIENT GLOBAL IMPRESSION OF IMPROVEMENT (PGI-I) SCALE

#### Patient Global Impression of Severity (PGI-S) Scale

Check the one number that best describes how your urinary tract condition is now.

- 1. Normal
- 2. Mild
- 3. Moderate
- 4. Severe

#### Patient Global Impression of Improvement (PGI-I) Scale

Check the one number that best describes how your urinary tract condition is now, compared with how it was before you began taking medication in this study.

- 1. Very much better
- 2. Much better
- 3. A little better
- 4. No change
- 5. A little worse
- 6. Much worse
- 7. Very much worse

Protocol: GTx-024 as a Treatment for Stress Urinary
Incontinence in Women: A Proof of Concept Study

Compound Incontinence in Women: A Proof of Concept Study

Compound No.: GTx-024 Author:

# 3. APPENDIX C: URINARY DISTRESS INVENTORY (UDI-6) AND INCONTINENCE IMPACT QUESTIONNAIRE (IIQ-7)

#### **Urinary Distress Inventory (UDI-6)**

- 1. Do you experience, and, if so, how much are you bothered by frequent urination?

  Not at all **0** Slightly **1** Moderately **3** Greatly**4**
- 2. Do you experience, and, if so, how much are you bothered by urine leakage related to the feeling of urgency?

Not at all **0** Slightly **1** Moderately **3** Greatly**4** 

3. Do you experience, and, if so, how much are you bothered by urine leakage related to physical activity, coughing, or sneezing?

Not at all **0** Slightly **1** Moderately **3** Greatly **4** 

4. Do you experience, and, if so, how much are you bothered by small amounts of urine leakage (drops)?

Not at all 0 Slightly 1 Moderately 3 Greatly4

5. Do you experience, and, if so, how much are you bothered by difficulty emptying your bladder?

Not at all 0 Slightly 1 Moderately 3 Greatly4

6. Do you experience, and, if so, how much are you bothered by pain or discomfort in the lower

abdominal or genital area?

Not at all 0 Slightly 1 Moderately 3 Greatly4

Protocol: GTx-024 as a Treatment for Stress Urinary
Incontinence in Women: A Proof of Concept Study

Compound No.: GTx-024
Author:

### **Incontinence Impact Questionnaire (IIQ-7)**

| 7. Has urine leakage affected your ability to do household chores (cooking, cleaning, laundry, etc)? | | | |
|---|---|---|---|
| <b>3</b> · | Slightly 1 | Moderately 3 | Greatly <b>4</b> |
| 8. Has urine leakaç<br>other exercise? | ge affected you | ur physical recreation | n such as walking, swimming, or |
| | Slightly 1 | Moderately 3 | Greatly <b>4</b> |
| - | • | ur entertainment acti<br><i>Moderately</i> <b>3</b> | vities (movies, concerts, etc.)? <i>Greatly</i> 4 |
| 10. Has urine leaka | age affected ye | our ability to travel by | y car or bus more than 30 minutes |
| | Slightly 1 | Moderately 3 | Greatly <b>4</b> |
| | | our participation in so<br><i>Moderately</i> <b>3</b> | ocial activities outside your house?<br><i>Greatly</i> <b>4</b> |
| | • | our emotional health<br><i>Moderately</i> <b>3</b> | (nervousness, depression, etc.)? <i>Greatly</i> <b>4</b> |
| | | our feeling frustrated<br><i>Moderately</i> <b>3</b> | |
| 14. Total Score for | UDI-6= | | |
| 15. Total Score for | IIQ-7= | | |

Protocol: GTx-024 as a Treatment for Stress Urinary
Incontinence in Women: A Proof of Concept Study

Compound No.: GTx-024
Author: \_\_\_\_\_

## 4. APPENDIX D: FEMALE SEXUAL FUNCTION INDEX (FSFI)

| Female Sexual Function Index (FSFI) | |
|---|---|
| Name | Date |
| INSTRUCTIONS: These questions ask about | your sexual feelings and responses during the |
| past 4 weeks. Please answer the following que | estions as honestly and clearly as possible. Your |
| responses will be kept completely confidential. | . In answering these questions the following |
| definitions apply: | |
| <u>Sexual activity</u> can include caressing, f | foreplay, masturbation and vaginal intercourse. |
| <u>Sexual intercourse</u> is defined as penile | penetration (entry) of the vagina. |
| <u>Sexual stimulation</u> includes situations I | like foreplay with a partner, self-stimulation |
| (masturbation), or sexual fantasy. | |
| CHECK <u>ONLY</u> ONE BOX PER QUESTION. | |
| Sexual desire or interest is a feeling that include | des wanting to have a sexual experience, feeling |
| receptive to a partner's sexual initiation, and th | ninking or fantasizing about having sex. |
| Over the past 4 weeks, how <b>often</b> did you for | eel sexual desire or interest? |
| ☐Almost always or always | |
| ☐Most times (more than half the time) | |
| ☐Sometimes (about half the time) | |
| ☐A few times (less than half the time) | |
| ☐Almost never or never | |
| 2. Over the past 4 weeks, how would you rate | your level (degree) of sexual desire |
| or interest? | |
| ☐Very high | |
| ∐High | |
| ☐Moderate | |
| □Low | |

| Protocol: GTx-024 as a Treatment for Stress Urinary Incontinence in Women: A Proof of Concept Study | Compound No.: GTx-024<br>Author: |
|---|---|
| ☐Very low or none at all | |
| Sexual arousal is a feeling that includes both physical and ment | al aspects of sexual excitement. |
| It may include feelings of warmth or tingling in the genitals, lubri | · |
| contractions. | , , , , |
| 3. Over the past 4 weeks, how <b>often</b> did you feel sexually arous | sed ("turned on") |
| during sexual activity or intercourse? | , |
| ☐No sexual activity | |
| ☐Almost always or always | |
| ☐Most times (more than half the time) | |
| ☐Sometimes (about half the time) | |
| ☐A few times (less than half the time) | |
| ☐Almost never | |
| 4. Over the past 4 weeks, how would you rate your <b>level</b> of sext | ual arousal ("turn |
| on") during sexual activity or intercourse? | |
| ☐No sexual activity | |
| ☐Very high | |
| ☐High | |
| ☐Moderate | |
| □Low | |
| ☐Very low or none at all | |
| 5. Over the past 4 weeks, how <b>confident</b> were you about become | ming sexually |
| aroused during sexual activity or intercourse? | |
| ☐No sexual activity | |
| ☐Very high confidence | |
| ☐High confidence | |
| ☐Moderate confidence | |
| Low confidence | |
| ☐Very low or no confidence | |
| 6. Over the past 4 weeks, how often have you been satisfied w | ith your arousal |
| (excitement) during sexual activity or intercourse? | |
| ☐No sexual activity | |
| ☐Almost always or always | |

| Protocol: GTx-024 as a Treatment for Stress Urinary Incontinence in Women: A Proof of Concept Study | Compound No.: GTx-024<br>Author: |
|---|---|
| ☐Most times (more than half the time) | |
| Sometimes (about half the time) | |
| ☐A few times (less than half the time) | |
| Almost never or never | |
| 7. Over the past 4 weeks, how <b>often</b> did you become lubricated | ("wet") durina |
| sexual activity or intercourse? | , 3 |
| ☐No sexual activity | |
| <br>∏Almost always or always | |
| ☐Most times (more than half the time) | |
| ☐Sometimes (about half the time) | |
| ☐A few times (less than half the time) | |
| ☐Almost never or never | |
| 8. Over the past 4 weeks, how <b>difficult</b> was it to become lubrical | ated ("wet") during |
| sexual activity or intercourse? | |
| ☐No sexual activity | |
| Extremely difficult or impossible | |
| □Very difficult | |
| ☐Difficult | |
| ☐Slightly difficult | |
| ☐Not difficult | |
| 9. Over the past 4 weeks, how often did you maintain your lubr | ication ("wetness") |
| until completion of sexual activity or intercourse? | |
| ☐No sexual activity | |
| ☐Almost always or always | |
| ☐Most times (more than half the time) | |
| ☐Sometimes (about half the time) | |
| ☐A few times (less than half the time) | |
| ☐Almost never or never | |
| 10. Over the past 4 weeks, how difficult was it to maintain your lubrication | |
| ("wetness") until completion of sexual activity or intercourse? | |
| ☐No sexual activity | |
| ☐Extremely difficult or impossible | |

| Protocol: GTx-024 as a Treatment for Stress Urinary Incontinence in Women: A Proof of Concept Study | Compound No.: GTx-024<br>Author: |
|---|---|
| ☐Very difficult | |
| ☐Difficult | |
| ☐Slightly difficult | |
| ☐Not difficult | |
| 11. Over the past 4 weeks, when you had sexual stimulation or | intercourse, how |
| often did you reach orgasm (climax)? | , |
| ☐No sexual activity | |
| ☐Almost always or always | |
| ☐Most times (more than half the time) | |
| Sometimes (about half the time) | |
| ☐A few times (less than half the time) | |
| ☐Almost never or never | |
| 12. Over the past 4 weeks, when you had sexual stimulation or | intercourse, how |
| difficult was it for you to reach orgasm (climax)? | |
| ☐No sexual activity | |
| ☐Extremely difficult or impossible | |
| ☐Very difficult | |
| Difficult | |
| ☐Slightly difficult | |
| ☐Not difficult | |
| 13. Over the past 4 weeks, how <b>satisfied</b> were you with your at | pility to reach orgasm |
| (climax) during sexual activity or intercourse? | |
| □No sexual activity | |
| ☐Very satisfied | |
| ☐Moderately satisfied | |
| About equally satisfied and dissatisfied | |
| ☐Moderately dissatisfied | |
| ☐Very dissatisfied | |
| 14. Over the past 4 weeks, how <b>satisfied</b> have you been with the amount of | |
| emotional closeness during sexual activity between you and your partner? | |

| Protocol: GTx-024 as a Treatment for Stress Urinary Incontinence in Women: A Proof of Concept Study | Compound No.: GTx-024<br>Author: |
|---|---|
| ☐Very satisfied | |
| ☐ Moderately satisfied | |
| ☐About equally satisfied and dissatisfied | |
| ☐ Moderately dissatisfied | |
| ☐Very dissatisfied | |
| 15. Over the past 4 weeks, how <b>satisfied</b> have you been with y | our sexual |
| relationship with your partner? | |
| □Very satisfied | |
| ☐ Moderately satisfied | |
| ☐About equally satisfied and dissatisfied | |
| ☐ Moderately dissatisfied | |
| ☐Very dissatisfied | |
| 16. Over the past 4 weeks, how <b>satisfied</b> have you been with y | our overall sexual life? |
| □Very satisfied | |
| ☐Moderately satisfied | |
| ☐About equally satisfied and dissatisfied | |
| ☐Moderately dissatisfied | |
| ☐Very dissatisfied | |
| _ , | |
| 17. Over the past 4 weeks, how <b>often</b> did you experience disco | mfort or pain during |
| vaginal penetration? | |
| ☐Did not attempt intercourse | |
| ☐Almost always or always | |
| ☐Most times (more than half the time) | |
| ☐Sometimes (about half the time) | |
| ☐A few times (less than half the time) | |
| ☐Almost never or never | |
| 18. Over the past 4 weeks, how often did you experience disco | mfort or pain following |
| vaginal penetration? | |
| ☐Did not attempt intercourse | |
| ☐Almost always or always | |
| ☐Most times (more than half the time) | |

| Protocol: GTx-024 as a Treatment for Stress Urinary Incontinence in Women: A Proof of Concept Study | Compound No.: GTx-024<br>Author: |
|---|---|
| ☐Sometimes (about half the time) ☐A few times (less than half the time) | |
| ☐Almost never or never 19.Over the past 4 weeks, how would you rate your <b>level</b> (degree) of discomfort or | |
| pain during or following vaginal penetration? | |
| ☐Did not attempt intercourse | ☐Did not attempt intercourse |
| ☐Very high | |
| □High | □High |
| ☐Moderate | |
| □Low | |
| ☐Very low or none at all | |
| Thank you for completing this questionnaire | |

GTx, Inc. SUI Protocol; Version 1.0

Protocol: GTx-024 as a Treatment for Stress Urinary
Incontinence in Women: A Proof of Concept Study

Compound No.: GTx-024
Author: \_\_\_\_\_\_

Study ID: \_\_\_\_\_

#### 5. APPENDIX E: VOIDING DIARY

**VOIDING DIARY** 

Wake Time: \_\_\_\_\_

ΑP

A P

ΑP

ΑP

ΑP

ΑP

| Bed Time: | | | | | | Date (m/d/y): | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time | Fluid Intake<br>(ounces) | Urine Amount<br>cc's/ml's or<br>ounces (oz) | first give th<br>"score" i<br>column th<br>you think it<br>urge incon<br>both in th | f you leak,<br>se episode a<br>n the first<br>en circle if<br>is stress or<br>tinence, or<br>ne second<br>umn) | Urgency | Pad<br>Replaced | Bowel Movement | Pelvic and/or<br>Bladder/Urinar<br>y Related Pain | Vaginal<br>discharge<br>color | Vaginal<br>discharge<br>amount |
| <b>A:</b> a.m.<br><b>P</b> : p.m. | | Amount Voided | 0: None<br>1: Mild<br>5: Mod.<br>10: Severe | <b>U</b> : Urge | 0: None<br>1: Mild<br>5: Mod.<br>10: Severe | 1: Tissue<br>2: Pantiliner<br>3: Thick Pad<br>4: Diaper | C: Constipated D: Diarrhea | 1: Mild<br>5: Mod<br>10: Severe | discharge<br>1: red<br>2: brown | 1: Spotting<br>2: dime size<br>3: quarter size<br>5: more than<br>quarter size |
| 5:00 AM | | | | S U | | | | | jo | |
| ΑP | | | | S U | | | | | | |
| ΑP | | | | S U | | | | | | |
| ΑP | | | | S U | | | | | | |
| ΑP | | | | S U | | | | | | |
| ΑP | | | | S U | | | | | | |
| ΑP | | | | S U | | | | | | |
| ΑP | | | | S U | | | | | | |
| ΑP | | | | S U | | | | | | |
| ΑP | | | | S U | | | | | | |

S U S U

S U

S U

S U

S U

S U